Replication of the ISAR-REACT 5 Trial in Healthcare Data Claims

NCT 01944800

August 3, 2021

#### 1. RCT Details

This section provides a high-level overview of the RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Ticagrelor or Prasugrel in Patients with Acute Coronary Syndromes (ISAR-REACT 5 trial)

#### 1.2 Intended aim(s)

To compare ticagrelor (180-mg loading dose, 90 mg twice daily thereafter) and prasugrel (60-mg loading dose, 10 mg daily thereafter) for the prevention of cardiovascular events in patients admitted to the hospital with an acute coronary syndrome, with or without ST-segment elevation, who were scheduled to undergo coronary angiography.

#### 1.3 Primary endpoint for replication and RCT finding

The primary outcome was composite of death, myocardial infarction, or stroke at 1 year after randomization

#### 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

Assuming an incidence of 10.0% in ticagrelor users and 12.9% in prasugrel users, 1,895 patients would be required for each group to achieve 80% power to detect a relative risk reduction of 22.5% in the rate of the primary outcome in the ticagrelor group as compared with the prasugrel group, using a two-sided alpha of 0.05.

#### 1.5 Primary trial estimate targeted for replication

HR = 1.36 (95% CI 1.09–1.70) comparing ticagrelor to prasugrel (Schupke et al., 2019)

#### 2. Person responsible for implementation of replication in Aetion

Dureshahwar Jawaid, MPH implemented the study design in the Aetion Evidence Platform. She is not responsible for the validity of the design and analytic choices. All implementation steps are recorded, and the implementation history is archived in the platform.

### 3. Data Source(s)

Optum, MarketScan

#### 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.



#### 5. Cohort Identification

#### 5.1 Cohort Summary

This study will involve a new user, parallel group, retrospective cohort study design comparing ticagrelor 90 mg twice daily to prasugrel 10 mg daily. The patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of ticagrelor or prasugrel (index date). We will restrict the analyses to patients with an acute coronary syndrome, with or without ST-segment elevation, who were scheduled to undergo coronary angiography.

#### 5.2 <u>Important steps for cohort formation</u>

New use of ticagrelor, exposure, and prasugrel comparator, is defined as no use of either therapy in 180 days prior to index date.

#### 5.2.1 Eligible cohort entry dates

Market availability of ticagrelor in the U.S. started on 2011-07-20.

- For Marketscan: 2011-07-20 to 2018-12-31 (end of data availability).
- For Optum: 2011-07-20 to 2020-03-31 (end of data availability).
- 5.2.2 Specify <u>inclusion/exclusion</u> criteria for cohort entry and define the index date. Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

#### 5.3 Flowchart of the study cohort assembly

| | Optum | Optum | | |
|---|---|---|---|---|
| | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients |
| All patients | | 78,779,380 | | 200,203,908 |
| Parent: Did not meet cohort entry criteria | 78,582,029 | 197,351 | -199978288 | 225,620 |
| Parent: Excluded due to insufficient enrollment | -27,693 | 169,658 | -56919 | 168,701 |
| Parent: Inclusion # 1.2.3 | -7,584 | 162,074 | -17110 | 151,591 |

| Parent: Excluded based on Start of Prasgurel 10mg OR Ticagrelor 90mg | -139,539 | 22,535 | -122209 | 29,382 |
|---|---|---|---|---|
| Parent: Excluded based on Exclusion # 13 - PCI | -1,511 | 21,024 | -1228 | 28,154 |
| Parent: Excluded based on Enrollment with allowed gap | -16 | 21,008 | -25 | 28,129 |
| Parent: Final cohort | | 21,008 | | 28,129 |
| Did not meet cohort entry criteria | 0 | 21,008 | 0 | 28,129 |
| Excluded due to insufficient enrollment | 0 | 21,008 | 0 | 28,129 |
| Excluded due to prior use of referent | -325 | 20,683 | -372 | 27,757 |
| Excluded due to prior use of exposure | -341 | 20,342 | -535 | 27,222 |
| Excluded because patient qualified in >1 exposure category | -5 | 20,337 | -3 | 27,219 |
| Excluded based on Inclusion # 2 - Age ≥ 18 | 0 | 20,337 | 0 | 27,219 |
| Excluded based on Exclusion # 2 - history of stroke or TIA | -6,788 | 13,549 | -6784 | 20,435 |
| Excluded based on Exclusion # 3 - intracranial neoplasm, intracranial AVM, intracranial aneurysm | -15 | 13,534 | -11 | 20,424 |
| Excluded based on Exclusion # 4 - Active bleeding | -446 | 13,088 | -595 | 19,829 |
| Excluded based on Exclusion # 6 - Thrombocytopenia | -269 | 12,819 | -261 | 19,568 |
| Excluded based on Exclusion # 7 - Anemia | -1,033 | 11,786 | -891 | 18,677 |
| Excluded based on Exclusion # 10 - chronic renal insufficiency | -38 | 11,748 | -37 | 18,640 |
| Excluded based on Exclusion # 11 - Moderate/severe hepatic dysfunction | -544 | 11,204 | -578 | 18,062 |
| Excluded based on Exclusion # 12 - Increased risk of bradycardia events | -342 | 10,862 | -413 | 17,649 |
| Excluded based on Exclusion # 14 - CCI ≥ 10 | -24 | 10,838 | -8 | 17,641 |
| Excluded based on Exclusion # 15 - Concomitant therapy with | | | | |
| strong CYP3A inhibitors/inducers | -28 | 10,810 | -53 | 17,588 |
| Excluded based on Exclusion # 19 - Pregnancy | -3 | 10,807 | -6 | 17,582 |
| Final cohort | | 10,807 | | 17,582 |

prior 6 months.

#### 6.2 <u>Preliminary covariates:</u>

- Age
- Sex

#### 6. Variables

# 6.1 <u>Exposure-related</u> <u>variables:</u>

#### Study drug:

The study exposure of interest is initiation of ticagrelor. Initiation will be defined as starting treatment with ticagrelor or a comparator drug with no prior use of the corresponding drug in the past 6 months (washout period).

#### Comparator agents:

New initiators of prasugrel 10 mg, defined by no use of ticagrelor or prasugrel in the • Combined Comorbidity Index (CCI), measured over the default baseline covariate assessment period, defined as 180 days prior to and including index date

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (**Appendix B**).

#### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Primary effectiveness outcomes of interest (definitions provided in **Appendix A**):

- Primary outcome: composite of death, myocardial infarction, or stroke at 1 year after randomization
- Secondary outcomes:
  - Individual components:
  - Hospital admission for MI
  - Hospital admission for stroke
  - Death

#### Safety outcomes of interest:

1. Major bleeding

#### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real-world databases is expected to be much worse than in the trial, the AT analysis is the **primary** analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analyses, the follow-up will start the day after initiation of ticagrelor and comparator and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,

Effectiveness research with Real World Data to support FDA's regulatory decision making

- End of the study period,
- Measured death event occurs,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (ticagrelor and comparator) plus a defined grace period (i.e., 30 days after the end of the last prescription's days' supply in main analyses).
- The date of augmentation or switching from exposure to comparator or vice versa
- The date of augmentation/switching from exposure or comparator to clopidogrel, measured as the initiation of clopidogrel starting from 1 day after cohort entry date
  - o A dosage change on the index treatment does not fulfill this criterion
  - o An added treatment that is not part of the exposure or comparator group does not fulfill this criterion

For the ITT analyses, the censoring based on the augmentation/switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

#### 7. Initial Feasibility Analysis

#### Aetion report links:

<u>Optum:</u> https://bwh-dope.aetion.com/projects/details/1740/rwrs/71503 <u>Marketscan:</u> https://bwh-dope.aetion.com/projects/details/1739/rwrs/71505

Date conducted: 06/11/2021

Complete Aetion feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

#### • Report patient characteristics by treatment group

| | Optum | | | | | |
|---|---|---|---|---|---|---|
| Variable | Exposure -<br>Ticagrelor<br>(90 mg) | Exposure -<br>Prasugrel<br>(10 mg) | Difference | Exposure -<br>Ticagrelor<br>(90 mg) | Exposure -<br>Prasugrel<br>(10 mg) | Difference |
| Number of patients | 6,722 | 4,085 | - (-, -) | 9,025 | 8,557 | - (-, -) |
| Age | | | | | | |
| mean (sd) | 63.60 (11.12) | 59.90<br>(10.02) | 3.70 (3.29,<br>4.11) | 58.41 (9.83) | 56.88<br>(8.90) | 1.54 (1.26,<br>1.81) |
| median [IQR] | 64.00 [56.00,<br>71.00] | 60.00<br>[53.00,<br>67.00] | - (-, -) | 59.00 [52.00,<br>63.00] | 58.00<br>[51.00,<br>63.00] | - (-, -) |
| Gender | | | | | | |
| 1 - Male; n (%) | 4,796<br>(71.3%) | 3,152<br>(77.2%) | -5.8% (-<br>7.5%, -<br>4.1%) | 6,790 (75.2%) | 6,835<br>(79.9%) | -4.6% (-<br>5.9%, -<br>3.4%) |
| 2 - Female; n (%) | 1,925<br>(28.6%) | 933<br>(22.8%) | 5.8%<br>(4.1%,<br>7.5%) | 2,235 (24.8%) | 1,722<br>(20.1%) | 4.6%<br>(3.4%,<br>5.9%) |
| CCI (180 days)- ICD9 and ICD10 | | | | | | |
| mean (sd) | 1.51 (1.96) | 0.93 (1.74) | 0.58 (0.51,<br>0.65) | 0.74 (1.54) | 0.50 (1.43) | 0.24 (0.19,<br>0.28) |
| median [IQR] | 1.00 [0.00,<br>3.00] | 1.00 [0.00,<br>2.00] | - (-, -) | 0.00 [0.00,<br>2.00] | 0.00 [-1.00,<br>1.00] | - (-, -) |

### • Report summary parameters of study population

| FEASIBILITY- FOR STUDY OUTCOME | | |
|-------------------------------------------------|--------|------------|
| | Optum | Marketscan |
| Variable | Value | Value |
| Number of patients in full cohort | 10,807 | 17,582 |
| Number of patients dropped as incomplete cases | 0 | 0 |
| Number of patients that did not begin follow-up | 3 | 5 |

| Number of patients in analytic cohort | 10,804 | 17,577 |
|---|---|---|
| Number of events | 777 | 1063 |
| Number of person-years | 7,415.55 | 13,945.70 |
| Number of patients in group: Exposure - Ticagrelor (90 mg) | 6,719 | 9,021 |
| Number of patients in group: Exposure - Prasugrel (10 mg) | 4,085 | 8,556 |
| Risk per 1,000 patients | 71.92 | 60.48 |
| Rate per 1,000 person-years | 104.78 | 76.22 |

### • Report median follow-up time by treatment group

| <u>, </u> | 1 1 1 | |
|---|---|---|
| MEDIAN FOLLOW-UP TIME FOR STUDY OUTCOME | | |
| Median Follow-Up Time (Days) [IQR] | | |
| Optum Marketscan | | |
| Patient Group Median Follow-Up Time (Days) [IQR] Median Follow-Up Time (Days) [IQR] | | |
| <b>Overall Patient Population</b> 196 [58, 391] 249 [91, 420] | | |
| <b>Referent</b> 172 [58, 386] 230 [85, 412] | | |
| Exposure | 232 [81, 403] | 273 [109, 433] |

### • Report reasons for censoring in the overall study population

| CENSORING REASONS FOR STUDY OUTCOME | | |
|-------------------------------------|------------|------------|
| Optum Marketscan | | |
| Overall | | |
| Outcome | 368 (3.4%) | 516 (2.9%) |

Effectiveness research with Real World Data to support FDA's regulatory decision making

| Death | 0 (0.0%) | 0 (0.0%) |
|---|---|---|
| Start of an additional exposure | 179 (1.7%) | 331 (1.9%) |
| End of index exposure | 4,994 (46.2%) | 8,242 (46.9%) |
| Specified date reached | 412 (3.8%) | 734 (4.2%) |
| End of patient data | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 1,873 (17.3%) | 4,889 (27.8%) |
| Switch to clopidogrel + Nursing home admission | 2,978 (27.6%) | 2,865 (16.3%) |

• Report overall risk of the primary outcome.

| | Optum | Marketscan | Pooled |
|-------------------------|-------|------------|--------|
| Risk per 1,000 patients | 71.92 | 60.48 | 64.81 |

#### 8. Initial Power Assessment

#### Aetion report links:

Optum: https://bwh-dope.aetion.com/projects/details/1740/rwrs/71504 Marketscan: https://bwh-dope.aetion.com/projects/details/1739/rwrs/71508

Date conducted: 06/11/2021

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

• Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.

### Pooled

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 24,266 |
| Reference | 12,133 |
| Exposed | 12,133 |
| Risk per 1,000 patients | 64.81 |
| Desired HR from RCT | 1.36 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 1572.67946 |
| Power | 0.999982406 |

### Marketscan

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 16,164 |
| Reference | 8,082 |
| Exposed | 8,082 |
| Risk per 1,000 patients | 60.48 |
| Desired HR from RCT | 1.36 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 977.59872 |
| Power | 0.997793559 |

Optum

Effectiveness research with Real World Data to support FDA's regulatory decision making

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 8,102 |
| Reference | 4,051 |
| Exposed | 4,051 |
| Risk per 1,000 patients | 71.92 |
| Desired HR from RCT | 1.36 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 582.69584 |
| Power | 0.960047459 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Date reviewed: |
|-------------------------|----------------|
| Reviewed by FDA: | Date reviewed: |
| Reasons for stopping | |
| analysis (if required): | |

#### 9. Balance Assessment

Aetion report name:

Optum: <a href="https://bwh-dope.aetion.com/projects/details/1740/rwrs/71506">https://bwh-dope.aetion.com/projects/details/1740/rwrs/71506</a>
Marketscan: <a href="https://bwh-dope.aetion.com/projects/details/1739/rwrs/71510">https://bwh-dope.aetion.com/projects/details/1739/rwrs/71510</a>

Date conducted: 06/10/2021

After review of initial feasibility and power analyses, complete creation of the remaining covariates from Section 6.2. Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates.

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

• Report covariate balance after matching.

Note- For Table 1, please refer to Appendix B.

Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy Outcome | 0 (0.00%) | 0 (0.00%) | 0 (0.00%) |
| Death | 45 (0.31%) | 17 (0.23%) | 28 (0.38%) |
| Start of an additional exposure | 307 (2.10%) | 248 (3.40%) | 59 (0.81%) |
| End of index exposure | 8,472 (58.03%) | 4,309 (59.03%) | 4,163 (57.03%) |
| Specified date reached | 602 (4.12%) | 245 (3.36%) | 357 (4.89%) |
| End of patient enrollment | 3,773 (25.84%) | 1,714 (23.48%) | 2,059 (28.21%) |
| Switch to clopidogrel + Nursing home admission | 1,401 (9.60%) | 767 (10.51%) | 634 (8.68%) |

• Report follow-up time by treatment group.

| Median Follow-Up Time (Days) [IQR] | | |
|------------------------------------|--------------|--------------|
| Patient Group Optum Marketscan | | |
| Overall Patient Population | 208 [58-395] | 259 [99-430] |
| Referent | 178 [58-391] | 241 [88-419] |

| Exposure | 229 [80-402] | 286 [112-445] |
|----------|--------------|---------------|
| · | | |

#### **10. Final Power Assessment**

Date conducted: 06/10/2021

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8.

#### Pooled

| 1 00100 | |
|----------------------------|-------------|
| Superiority Analysis | |
| Number of patients matched | 14,600 |
| Reference | 7,300 |
| Exposed | 7,300 |
| Risk per 1,000 patients | 65.52 |
| Desired HR from RCT | 1.36 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 956.592 |
| Power | 0.997405863 |

Marketscan

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 9,604 |
| Reference | 4,802 |
| Exposed | 4,802 |
| Risk per 1,000 patients | 61.61 |
| Desired HR from RCT | 1.36 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 591.70244 |
| Power | 0.962446362 |

Optum

Effectiveness research with Real World Data to support FDA's regulatory decision making

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 4,996 |
| Reference | 2,498 |
| Exposed | 2,498 |
| Risk per 1,000 patients | 71.92 |
| Desired HR from RCT | 1.36 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 359.31232 |
| Power | 0.830035796 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Date reviewed: |
|-------------------------|----------------|
| Reviewed by FDA: | Date reviewed: |
| Reasons for stopping | |
| analysis (if required): | |

#### 11. Study Confidence and Concerns

<u>Deadline for voting on study confidence and listing concerns:</u>

Date votes and concerns are summarized:

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the success of the RWD study in the <u>Google Form</u>. This form also provides space for reviewers to list any concerns that they feel may

contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the individual respondent.

• After the deadline for voting has passed, provide the distribution of responses and summarize all concerns here.

#### 12. Register study protocol on clinicalTrials.gov

#### Date conducted:

• Register the study on <u>clinicalTrials.gov</u> and upload this document.

#### 13. Comparative Analyses

Aetion report name:

Date conducted:

- 13.1 For primary analysis:
- 13.2 For sensitivity analyses:

#### 14. Requested Results

#### 14.1 Table 1: Baseline characteristics before and after adjustment

| Variable | Before adjustment | | After adjustment | | | |
|---|---|---|---|---|---|---|
| | Referent | Exposure | Std. diff. | Referent | Exposure | Std. diff. |
| Number of patients | | | - | | | - |
| Age categories | | | | | | |

### 14.2 <u>Table 2: Follow-up time</u>

| Patient Group Median Follow-Up Time (Days) [IQR] |
|--------------------------------------------------|
| Overall Patient Population |
| Referent |
| Exposure |

#### 14.3 <u>Table 3: Censoring events</u>

| | Overall | Referent | Exposure |
|---------------------------------|---------|----------|----------|
| Outcome | | | |
| Death | | | |
| Start of an additional exposure | | | |
| End of index exposure | | | |
| Specified date reached | | | |
| End of patient data | | | |
| End of patient enrollment | | | |

#### 14.4 <u>Table 4: Results from primary analyses;</u>

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Analysis 1 | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

### 14.5 <u>Table 5: Results from secondary analyses;</u>

Effectiveness research with Real World Data to support FDA's regulatory decision making

#### 15. References

Schupke S., Neumann F., Menichelli M., et al. Ticagrelor or Prasugrel in Patients with Acute Coronary Syndromes. N Engl J Med. 2019; 381:1524-1534

Chow S, Shao J, Wang H. 2008. *Sample Size Calculations in Clinical Research*. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177

**NCT** 

Trial Name (with web links)

**ISAR-REACT 5** 

**Trial Name (with pdf links)** 

ISAR-REACT 5 NCT01944800

Therapeutic Area Cardiology/Vascular Diseases

<u>Study Batch</u> Antiplatelets

Brand NameBrilintaGeneric NameTicagrelor

<u>Sponsor</u> Deutsches Herzzentrum Muenchen

<u>Year</u> 2019

Measurable Endpoint The primary end point was the composite of

stroke, myocardial infarction, or death

<u>Exposure</u> Ticagrelor <u>Comparator</u> Prasugrel

Patients who were hospitalized for an acute coronary syndrome (ST-segment

<u>Population</u> elevation myocardial infarction, non-ST-segment elevation myocardial

infarction or unstable angina pectoris) with planned invasive strategy

<u>Trial Finding</u> HR = 1.36 (95% CI, 1.09 to 1.70)

<u>No. of Patients</u> 4,018 (2,012 in exposed arm)

80% power; 1895 patients in each group would be needed for the trial to detect

**Power** a relative risk

that was lower by 22.5% in the rate of the primary end point in the ticagrelor

group as compared with the prasugrel group

Coronary angiography

### Procedure codes any diagnosis position, inpatient and outpatient setting Source: https://www.cordis.com/content/dam/cordis/web/documents/fact-sheet/cordis-cardiology-reimbursement-fact-CPT 93451 performed Left heart catheterization including intraprocedural injection(s) for left ventriculography, imaging 93452 supervision and interpretation, when performed Combined right and left heart catheterization including intraprocedural injection(s) for left ventriculography, 93453 imaging supervision and interpretation, when performed 93454 Coronary angiography 93455 Coronary angiography with bypass grafts 93456 Coronary angiography with right heart catheterization 93457 Coronary angiography and bypass grafts, with right heart catheterization 93458 Coronary angiography with left heart catheterization 93459 Coronary angiography and bypass grafts, with left heart catheterization 93460 Coronary angiography with right and left heart catheterization 93461 Coronary angiography with bypass grafts, right and left heart catheterization 93563 Injection/imaging for coronary angiography with cath for congenital anomaly 93564 Injection/imaging for bypass graft angiography with cath for congenital anomaly 93565 Injection/imaging for left heart angiography with cath for congenital anomaly 93566 Injection/imaging for right heart angiography with cath for congenital anomaly Computed tomographic angiography, heart, coronary arteries and bypass grafts (when present), with 75574 contrast material, including 3D image postprocessing (including evaluation of cardiac structure and morphology, assessment of cardiac function, and evaluation of venous structures, if performed) ICD-9 PX 37.21 Right heart cardiac catheterization 37.22 Left heart cardiac catheterization 37.23 Combined right and left heart cardiac catheterization

| B21 | Fluoroscopy (heart) |
|---------|-----------------------------------------|
| B210xxx | Coronary Arterias Multiple |
| B211xxx | Coronary Arteries, Multiple |
| B212xxx | Coronary Artery Bypass Graft, Single |
| B213xxx | Coronary Artery Bypass Grafts, Multiple |
| B214xxx | Heart, Right |
| B215xxx | Heart, Left |
| B216xxx | Heart, Right and Left |
| B217xxx | Internal Mammary Bypass Graft, Right |
| B218xxx | Internal Mammary Bypass Graft, Left |
| B21Fxxx | Bypass Graft, Other |
| B22 | CT Scan (heart) |
| B221xxx | Coronary Arteries, Multiple |
| B223xxx | Coronary Artery Bypass Grafts, Multiple |
| B226xxx | Heart, Right and Left |
| B31 | Fluoroscopy (upper arteries) |
| B312xxx | Subclavian Artery, Left |
| B313xxx | Common Carotid Artery, Right |
| B314xxx | Common Carotid Artery, Left |
| B315xxx | Common Carotid Arteries, Bilateral |
| B316xxx | Internal Carotid Artery, Right |
| B317xxx | Internal Carotid Artery, Left |
| B318xxx | Internal Carotid Arteries, Bilateral |
| B319xxx | External Carotid Artery, Right |
| B31Bxxx | External Carotid Artery, Left |
| B31Cxxx | External Carotid Arteries, Bilateral |
| B32 | CT scan (upper arteries) |
| B325xxx | Common Carotid Arteries, Bilateral |
| B328xxx | Internal Carotid Arteries, Bilateral |
| | · |

Major bleeding exclusion criteria: 1 inpatient (any position) or 2 outpatient diagnosis (separated by 7-365 days)


| $\mathbf{r}$ | • | • |
|--------------|---|---|
| | • | |
| г | • | |

Procedure codes in any position, inpatient or outpatient setting


#### ICD-9 px codes:

| - |
|---|

### ICD-10 px codes:

027004Z (ICD10) Dilation of Coronary Artery, One Artery with Drug


#### Title

Pregnancy


| ICD-9 Px inpatient any position | |
|---|---|
| 72.0 | Low forceps operation |
| 72.1 | Low forceps operation with episiotomy |
| 72.2 | Mid forceps operation |
| 72.21 | Mid forceps operation with episiotomy |
| 72.29 | Other mid forceps operation |
| 72.3 | High forceps operation |
| 72.31 | High forceps operation with episiotomy |
| 72.39 | Other high forceps operation |
| 72.4 | Forceps rotation of fetal head |
| 72.5 | Breech extraction |
| 72.51 | Partial breech extraction with forceps to aftercoming head |
| 72.52 | Other partial breech extraction |
| 72.53 | Total breech extraction with forceps to aftercoming head |
| 72.54 | Other total breech extraction |
| 72.6 | Forceps application to aftercoming head |
| 72.7 | Vacuum extraction |
| 72.71 | Vacuum extraction with episiotomy |
| 72.79 | Other vacuum extraction |
| 72.8 | Other specified instrumental delivery |
| 72.9 | Unspecified instrumental delivery |
| 73.0 | Artificial rupture of membranes |
| 73.01 | Induction of labor by artificial rupture of membranes |
| 73.09 | Other artificial rupture of membranes |
| 73.1 | Other surgical induction of labor |
| 73.2 | Internal and combined version and extraction |
| 73.21 | Internal and combined version without extraction |
| 73.22 | Internal and combined version with extraction |
| 73.3 | Failed forceps |
| 73.4 | Medical induction of labor |
| 73.5 | Manually assisted delivery |

| 73.51 | Manual rotation of fetal head |
|-------|--------------------------------------------------|
| 73.59 | Other manually assisted delivery |
| 73.6 | Episiotomy |
| 73.8 | Operations on fetus to facilitate delivery |
| 73.9 | Other operations assisting delivery |
| 73.91 | External version assisting delivery |
| 73.92 | Replacement of prolapsed umbilical cord |
| 73.93 | Incision of cervix to assist delivery |
| 73.94 | Pubiotomy to assist delivery |
| 73.99 | Other operations assisting delivery |
| 74.0 | Classical cesarean section |
| 74.1 | Low cervical cesarean section |
| 74.2 | Extraperitoneal cesarean section |
| 74.3 | Removal of extratubal ectopic pregnancy |
| 74.4 | Cesarean section of other specified type |
| 74.9 | Cesarean section of unspecified type |
| 74.91 | Hysterotomy to terminate pregnancy |
| 74.99 | Other cesarean section of unspecified type |
| 75.4 | Manual removal of retained placenta |
| 75.5 | Repair of current obstetric laceration of uterus |
| 75.6 | Repair of other current obstetric laceration |
| 75.7 | Manual exploration of uterine cavity, postpartum |
| 75.9 | Other obstetric operations |







| | | Optum | | | Marketscan | | | Pooled | |
|---|---|---|---|---|---|---|---|---|---|
| | Ticagrelor | Prasugrel | St. Diff | Ticagrelor | Prasugrel | St. Diff | Ticagrelor | Prasugrel | St. Diff |
| Number of patients | 6,722 | 4,085 | | 9,025 | 8,557 | | 15,747 | 12,642 | |
| Quarter/Year of Cohort Entry Date | | | | | | | | | |
| Q3 2011; n (%) | 1 (0.0%) | 169 (4.1%) | -0.2924 | 2 (0.0%) | 478 (5.6%) | -0.3444 | 003 (0.0%) | 647 (5.1%) | -0.328 |
| Q4 2011; n (%) | 2 (0.0%) | 195 (4.8%) | -0.3176 | 19 (0.2%) | 644 (7.5%) | -0.3864 | 021 (0.1%) | 839 (6.6%) | -0.367 |
| Q1 2012; n (%) | 11 (0.2%) | 165 (4.0%) | -0.2674 | 51 (0.6%) | 695 (8.1%) | -0.3741 | 062 (0.4%) | 860 (6.8%) | -0.349 |
| Q2 2012; n (%) | 30 (0.4%) | 187 (4.6%) | -0.2715 | 104 (1.2%) | 607 (7.1%) | -0.2991 | 134 (0.9%) | 794 (6.3%) | -0.293 |
| Q3 2012; n (%) | 44 (0.7%) | 181 (4.4%) | -0.2363 | 142 (1.6%) | 621 (7.3%) | -0.2791 | 186 (1.2%) | 802 (6.3%) | -0.271 |
| Q4 2012; n (%) | 42 (0.6%) | 177 (4.3%) | -0.2411 | 177 (2.0%) | 557 (6.5%) | -0.2245 | 219 (1.4%) | 734 (5.8%) | -0.238 |
| Q1 2013; n (%) | 80 (1.2%) | 168 (4.1%) | -0.1813 | 172 (1.9%) | 373 (4.4%) | -0.1435 | 252 (1.6%) | 541 (4.3%) | -0.160 |
| Q2 2013; n (%) | 95 (1.4%) | 143 (3.5%) | -0.1362 | 196 (2.2%) | 302 (3.5%) | -0.0782 | 291 (1.8%) | 445 (3.5%) | -0.106 |
| Q3 2013; n (%) | 75 (1.1%) | 147 (3.6%) | -0.1656 | 255 (2.8%) | 376 (4.4%) | -0.0860 | 330 (2.1%) | 523 (4.1%) | -0.116 |
| Q4 2013; n (%) | 82 (1.2%) | 139 (3.4%) | -0.1472 | 275 (3.0%) | 315 (3.7%) | -0.0389 | 357 (2.3%) | 454 (3.6%) | -0.077 |
| Q1 2014; n (%) | 81 (1.2%) | 122 (3.0%) | -0.1258 | 245 (2.7%) | 296 (3.5%) | -0.0462 | 326 (2.1%) | 418 (3.3%) | -0.074 |
| Q2 2014; n (%) | 92 (1.4%) | 126 (3.1%) | -0.1148 | 319 (3.5%) | 301 (3.5%) | 0.0000 | 411 (2.6%) | 427 (3.4%) | -0.047 |
| Q3 2014; n (%) | 109 (1.6%) | 117 (2.9%) | -0.0877 | 399 (4.4%) | 312 (3.6%) | 0.0408 | 508 (3.2%) | 429 (3.4%) | -0.011 |
| Q4 2014; n (%) | 109 (1.6%) | 117 (2.9%) | -0.0877 | 430 (4.8%) | 297 (3.5%) | 0.0652 | 539 (3.4%) | 414 (3.3%) | 0.006 |
| Q1 2015; n (%) | 92 (1.4%) | 87 (2.1%) | -0.0534 | 335 (3.7%) | 190 (2.2%) | 0.0887 | 427 (2.7%) | 277 (2.2%) | 0.032 |
| Q2 2015; n (%) | 102 (1.5%) | 78 (1.9%) | -0.0309 | 354 (3.9%) | 166 (1.9%) | 0.1194 | 456 (2.9%) | 244 (1.9%) | 0.065 |
| Q3 2015; n (%) | 110 (1.6%) | 96 (2.4%) | -0.0572 | 436 (4.8%) | 191 (2.2%) | 0.1418 | 546 (3.5%) | 287 (2.3%) | 0.072 |
| Q4 2015; n (%) | 130 (1.9%) | 124 (3.0%) | -0.0712 | 483 (5.4%) | 234 (2.7%) | 0.1373 | 613 (3.9%) | 358 (2.8%) | 0.061 |
| Q1 2016; n (%) | 117 (1.7%) | 129 (3.2%) | -0.0971 | 462 (5.1%) | 247 (2.9%) | 0.1124 | 579 (3.7%) | 376 (3.0%) | 0.039 |
| Q1 2016; n (%) | 170 (2.5%) | 118 (2.9%) | -0.0247 | 497 (5.5%) | 231 (2.7%) | 0.1124 | 667 (4.2%) | 349 (2.8%) | 0.076 |
| Q2 2016; n (%) | 199 (3.0%) | 130 (3.2%) | -0.0115 | 534 (5.9%) | 232 (2.7%) | 0.1582 | 733 (4.7%) | 362 (2.9%) | 0.094 |
| Q3 2016; it (%) | 213 (3.2%) | 133 (3.3%) | -0.0056 | 576 (6.4%) | 225 (2.6%) | 0.1382 | 789 (5.0%) | 358 (2.8%) | 0.034 |
| Q4 2016, II (%)<br>Q1 2017; n (%) | 276 (4.1%) | · ' | 0.0713 | | · ' | 0.2104 | 800 (5.1%) | 271 (2.1%) | 0.114 |
| - / / / | | 113 (2.8%)<br>122 (3.0%) | 0.0713 | 524 (5.8%)<br>578 (6.4%) | 158 (1.8%)<br>162 (1.9%) | 0.2104 | 989 (6.3%) | 284 (2.2%) | 0.102 |
| Q2 2017; n (%) | 411 (6.1%) | . , | 0.1492 | 693 (7.7%) | | 0.2556 | 1,183 (7.5%) | 317 (2.5%) | 0.204 |
| Q3 2017; n (%) | 490 (7.3%) | 125 (3.1%) | 0.1900 | ` ' | 192 (2.2%) | 0.3034 | 1,334 (8.5%) | 276 (2.2%) | 0.231 |
| Q4 2017; n (%) | 578 (8.6%) | 122 (3.0%) | | 756 (8.4%) | 154 (1.8%) | 0.3034 | ' ' ' | 097 (0.8%) | 0.283 |
| Q1 2018; n (%) | 535 (8.0%) | 96 (2.4%) | 0.2543 | 11 (0.1%) | 1 (0.0%) | 0.0447 | 546 (3.5%) | 097 (0.8%) | 0.187 |
| Demographics | | | | | | | | | |
| Age<br>mean (sd) | 63.60 (11.12) | 59.90 (10.02) | 0.3496 | 58.41 (9.83) | 56.88 (8.90) | 0.1632 | 60.63 (10.40) | 57.86 (9.28) | 0.281 |
| median [IQR] | ` ' | 60.00 [53.00, 67.00] | 0.3779 | ` ' | 58.00 [51.00, 63.00] | 0.1032 | 61.13 (10.40) | 58.65 (9.28) | 0.251 |
| Gender without zero category- United | 64.00 [56.00, 71.00] | 60.00 [53.00, 67.00] | 0.3779 | 59.00 [52.00, 63.00] | 58.00 [51.00, 63.00] | 0.1000 | 01.13 (10.40) | 36.03 (3.26) | 0.232 |
| Males; n (%) | 4,796 (71.3%) | 3,152 (77.2%) | -0.1352 | 6,790 (75.2%) | 6,835 (79.9%) | -0.0054 | 11,586 (73.6%) | 9,987 (79.0%) | -0.127 |
| | 1,925 (28.6%) | 933 (22.8%) | 0.1332 | 2,235 (24.8%) | 1,722 (20.1%) | -0.0054 | 4,160 (26.4%) | 2,655 (21.0%) | 0.127 |
| Females; n (%)Missing; n (%) | 1,925 (28.6%) | 0 (0.0%) | #DIV/0! | 2,233 (24.6%) | 1,722 (20.1%) | -0.0034 | 4,100 (20.470) | 2,033 (21.070) | 0.127 |
| Region without zero category- United v3 (lumping missing | | 0 (0.070) | #514/0: | | | | | | |
| Northeast; n (%) | 732 (10.9%) | 300 (7.3%) | 0.1254 | 1,683 (18.6%) | 1,345 (15.7%) | 0.0770 | 2,415 (15.3%) | 1,645 (13.0%) | 0.066 |
| South; n (%) | 2,955 (44.0%) | 2,035 (49.8%) | -0.1164 | 3,993 (44.2%) | 3,705 (43.3%) | 0.0181 | 6,948 (44.1%) | 5,740 (45.4%) | -0.026 |
| Midwest; n (%) | 1,721 (25.6%) | 929 (22.7%) | 0.0678 | 2,321 (25.7%) | 2,089 (24.4%) | 0.0300 | 4,042 (25.7%) | 3,018 (23.9%) | 0.042 |
| West; n (%) | 1,314 (19.5%) | 821 (20.1%) | -0.0151 | 970 (10.7%) | 1,285 (15.0%) | -0.1288 | 2,284 (14.5%) | 2,106 (16.7%) | -0.061 |
| Metropolitan Statistical Area - Urban (any MSA) vs Rural | <u> </u> | 021 (20.1/0) | 0.0131 | J, U (10.7/0) | 1,203 (13.0/0) | 0.1200 | 2,207 (17.3/0) | 2,100 (10.770) | 5.001 |
| Urban; n (%) | (HOII WISA) | | | 6,388 (70.8%) | 6,604 (77.2%) | -0.1463 | 6,388 (70.8%) | 6,604 (77.2%) | -0.1463 |
| Rural; n (%) | | | | 710 (7.9%) | 207 (2.4%) | 0.2508 | 710 (7.9%) | 207 (2.4%) | 0.2508 |
| Unknown/Missing; n (%) | 1 | | | 1,927 (21.4%) | 1,746 (20.4%) | 0.0246 | 1,927 (21.4%) | 1,746 (20.4%) | 0.0246 |
| Commercial vs Medicare Advantage- Business Type Code | 1 | 1 | | -,52. (22.7/0) | _, (20.7/0) | | _,5, 70] | _, (20.470) | |
| COM = COMMERCIAL; n (%) | 3,343 (49.7%) | 2,633 (64.5%) | -0.3024 | | | | 3,343 (49.7%) | 2,633 (64.5%) | -0.3024 |
| MCR = MEDICARE; n (%) | 3,379 (50.3%) | 1,452 (35.5%) | 0.3024 | | | | 3,379 (50.3%) | 1,452 (35.5%) | 0.3024 |

| MCD = MEDICAID; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | | | | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
|---|---|---|---|---|---|---|---|---|---|
| NONE = NO BUSINESS LINE CODE (added in 2015); n (%) | | 0 (0.0%) | #DIV/0! | | | | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| UNK = UNKNOWN (added in 2015); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | | | | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Commercial vs Medicare Advantage- Data Type | , , | , , | | | | | , , | , , | |
| 1 - Fee For Service; n (%) | | | | 6,570 (72.8%) | 6,428 (75.1%) | -0.0524 | 6,570 (72.8%) | 6,428 (75.1%) | -0.0524 |
| 2 - Encounter; n (%) | | | | 732 (8.1%) | 757 (8.8%) | -0.0252 | 732 (8.1%) | 757 (8.8%) | -0.0252 |
| 3 - Medicare; n (%) | | | | 1,510 (16.7%) | 1,196 (14.0%) | 0.0750 | 1,510 (16.7%) | 1,196 (14.0%) | 0.0750 |
| 4 - Medicare Encounter; n (%) | | | | 213 (2.4%) | 176 (2.1%) | 0.0202 | 213 (2.4%) | 176 (2.1%) | 0.0202 |
| Lifestyle factors | | | | | | | | | |
| Obesity; n (%) | 1,853 (27.6%) | 1,014 (24.8%) | 0.0637 | 1,853 (20.5%) | 1,538 (18.0%) | 0.0634 | 3,706 (23.5%) | 2,552 (20.2%) | 0.080 |
| Overweight; n (%) | 480 (7.1%) | 194 (4.7%) | 0.1020 | 330 (3.7%) | 161 (1.9%) | 0.1093 | 810 (5.1%) | 355 (2.8%) | 0.118 |
| Smoking; n (%) | 3,323 (49.4%) | 1,925 (47.1%) | 0.0460 | 2,999 (33.2%) | 2,822 (33.0%) | 0.0043 | 6,322 (40.1%) | 4,747 (37.5%) | 0.053 |
| Alcohol abuse or dependence+Drug abuse or dependence ( | ( 377 (5.6%) | 168 (4.1%) | 0.0699 | 293 (3.2%) | 266 (3.1%) | 0.0057 | 670 (4.3%) | 434 (3.4%) | 0.047 |
| Diabetes-related conditions | | | | | | | | | |
| Diabetic retinopathy; n (%) | 138 (2.1%) | 60 (1.5%) | 0.0451 | 115 (1.3%) | 99 (1.2%) | 0.0090 | 253 (1.6%) | 159 (1.3%) | 0.025 |
| Occurrence of Diabetic Neuropathy v2 Copy; n (%) | 463 (6.9%) | 185 (4.5%) | 0.1037 | 318 (3.5%) | 249 (2.9%) | 0.0341 | 781 (5.0%) | 434 (3.4%) | 0.080 |
| Occurrence of diabetic nephropathy V3 with ICD10 Copy; n | | 132 (3.2%) | 0.1215 | 219 (2.4%) | 132 (1.5%) | 0.0651 | 605 (3.8%) | 264 (2.1%) | 0.101 |
| Hypoglycemia v2; n (%) | 21 (0.3%) | 36 (0.9%) | -0.0778 | 71 (0.8%) | 79 (0.9%) | -0.0109 | 092 (0.6%) | 115 (0.9%) | -0.035 |
| Hyperglycemia; n (%) | 527 (7.8%) | 318 (7.8%) | 0.0000 | 563 (6.2%) | 438 (5.1%) | 0.0477 | 1,090 (6.9%) | 756 (6.0%) | 0.037 |
| Disorders of fluid electrolyte and acid-base balance; n (%) | 968 (14.4%) | 461 (11.3%) | 0.0927 | 815 (9.0%) | 691 (8.1%) | 0.0322 | 1,783 (11.3%) | 1,152 (9.1%) | 0.073 |
| Hyperosmolar hyperglycemic nonketotic syndrome (HONK) | 21 (0.3%) | 12 (0.3%) | 0.0000 | 8 (0.1%) | 10 (0.1%) | 0.0000 | 029 (0.2%) | 022 (0.2%) | 0.000 |
| Diabetic Foot; n (%) | 57 (0.8%) | 27 (0.7%) | 0.0116 | 45 (0.5%) | 54 (0.6%) | -0.0135 | 102 (0.6%) | 081 (0.6%) | 0.000 |
| Skin infections v2; n (%) | 212 (3.2%) | 134 (3.3%) | -0.0056 | 265 (2.9%) | 261 (3.1%) | -0.0117 | 477 (3.0%) | 395 (3.1%) | -0.006 |
| Erectile dysfunction; n (%) | 198 (2.9%) | 141 (3.5%) | -0.0341 | 244 (2.7%) | 198 (2.3%) | 0.0256 | 442 (2.8%) | 339 (2.7%) | 0.006 |
| Diabetes with unspecified complication; n (%) | 231 (3.4%) | 84 (2.1%) | 0.0796 | 223 (2.5%) | 184 (2.2%) | 0.0198 | 454 (2.9%) | 268 (2.1%) | 0.051 |
| Diabetes mellitus without mention of complications; n (%) | | 1,403 (34.3%) | -0.0042 | 2,797 (31.0%) | 2,784 (32.5%) | -0.0322 | 5,087 (32.3%) | 4,187 (33.1%) | -0.017 |
| Diabetes with peripheral circulatory disorders+Gangrene+ | | 66 (1.6%) | 0.1207 | 125 (1.4%) | 97 (1.1%) | 0.0270 | 357 (2.3%) | 163 (1.3%) | 0.075 |
| Diabetes with other ophthalmic manifestations+Retinal de | <u> </u> | 14 (0.3%) | 0.0448 | 80 (0.9%) | 90 (1.1%) | -0.0201 | 123 (0.8%) | 104 (0.8%) | 0.000 |
| Cardiovascular-related conditions | | (2.2.7) | | | | | | , , | |
| Hypertension: 1 inpatient or 2 outpatient claims within 36 | 5,346 (79.5%) | 3,106 (76.0%) | 0.0842 | 6,673 (73.9%) | 5,846 (68.3%) | 0.1238 | 12,019 (76.3%) | 8,952 (70.8%) | 0.125 |
| Malignant hypertension; n (%) | 171 (2.5%) | 190 (4.7%) | -0.1183 | 2,791 (30.9%) | 4,225 (49.4%) | -0.3843 | 2,962 (18.8%) | 4,415 (34.9%) | -0.369 |
| Hyperlipidemia v2; n (%) | 5,379 (80.0%) | 3,348 (82.0%) | -0.0510 | 6,450 (71.5%) | 5,864 (68.5%) | 0.0655 | 11,829 (75.1%) | 9,212 (72.9%) | 0.050 |
| Acute MI; n (%) | 6,184 (92.0%) | 3,877 (94.9%) | -0.1174 | 8,521 (94.4%) | 8,293 (96.9%) | -0.1228 | 14,705 (93.4%) | 12,170 (96.3%) | -0.131 |
| ACS/unstable angina; n (%) | 2,766 (41.1%) | 1,553 (38.0%) | 0.0634 | 3,475 (38.5%) | 3,016 (35.2%) | 0.0684 | 6,241 (39.6%) | 4,569 (36.1%) | 0.072 |
| Old MI; n (%) | 952 (14.2%) | 510 (12.5%) | 0.0500 | 774 (8.6%) | 705 (8.2%) | 0.0144 | 1,726 (11.0%) | 1,215 (9.6%) | 0.046 |
| Stable angina; n (%) | 1,583 (23.5%) | 665 (16.3%) | 0.1811 | 1,561 (17.3%) | 1,077 (12.6%) | 0.1321 | 3,144 (20.0%) | 1,742 (13.8%) | 0.166 |
| Coronary atherosclerosis and other forms of chronic ischer | · · · · · · | 3,951 (96.7%) | -0.0322 | 8,365 (92.7%) | 7,850 (91.7%) | 0.0373 | 14,826 (94.2%) | 11,801 (93.3%) | 0.037 |
| Ischemic stroke (w and w/o mention of cerebral infarction | | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| TIA; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| Late effects of cerebrovascular disease; n (%) | 26 (0.4%) | 6 (0.1%) | 0.0601 | 9 (0.1%) | 9 (0.1%) | 0.0000 | 035 (0.2%) | 015 (0.1%) | 0.026 |
| Heart failure (CHF); n (%) | 1,300 (19.3%) | 634 (15.5%) | 0.1004 | 1,206 (13.4%) | 1,105 (12.9%) | 0.0148 | 2,506 (15.9%) | 1,739 (13.8%) | 0.059 |
| Peripheral Vascular Disease (PVD) or PVD Surgery v2; n (% | <u> </u> | 164 (4.0%) | 0.0706 | 250 (2.8%) | 232 (2.7%) | 0.0061 | 619 (3.9%) | 396 (3.1%) | 0.044 |
| Atrial fibrillation; n (%) | 541 (8.0%) | 252 (6.2%) | 0.0701 | 454 (5.0%) | 355 (4.1%) | 0.0432 | 995 (6.3%) | 607 (4.8%) | 0.066 |
| Other cardiac dysrhythmia; n (%) | 2,369 (35.2%) | 1,204 (29.5%) | 0.1221 | 2,553 (28.3%) | 2,010 (23.5%) | 0.1097 | 4,922 (31.3%) | 3,214 (25.4%) | 0.131 |
| Hemorrhagic stroke+Other cerebrovascular disease+Cereb | <u> </u> | 13 (0.3%) | 0.0448 | 28 (0.3%) | 14 (0.2%) | 0.0200 | 067 (0.4%) | 027 (0.2%) | 0.037 |
| Other atherosclerosis+Cardiac conduction disorders+Other | <del>- ' '</del> | 1,384 (33.9%) | 0.0917 | 2,672 (29.6%) | 2,323 (27.1%) | 0.0555 | 5,244 (33.3%) | 3,707 (29.3%) | 0.086 |
| Previous cardiac procedure (CABG or PTCA or Stent) + Hist | , | 4,012 (98.2%) | -0.0286 | 8,349 (92.5%) | 7,936 (92.7%) | -0.0076 | 14,924 (94.8%) | 11,948 (94.5%) | 0.013 |
| Kidney-related conditions | 5,575 (57.670) | -1,012 (30.2/0) | 3.3200 | 5,575 (52.570) | 7,330 (32.770) | 3.3070 | 2.,52. (54.070) | 22,5 :5 (54.576) | 5.515 |
| Occurrence of acute renal disease v2; n (%) | 533 (7.9%) | 227 (5.6%) | 0.0918 | 425 (4.7%) | 294 (3.4%) | 0.0660 | 958 (6.1%) | 521 (4.1%) | 0.091 |
| Occurrence of hypertensive nephropathy; n (%) | 543 (8.1%) | 212 (5.2%) | 0.1166 | 316 (3.5%) | 229 (2.7%) | 0.0462 | 859 (5.5%) | 441 (3.5%) | 0.097 |
| Occurrence of miscellaneous renal insufficiency v2; n (%) | <u> </u> | 187 (4.6%) | 0.0187 | 272 (3.0%) | 226 (2.6%) | 0.0242 | 610 (3.9%) | 413 (3.3%) | 0.032 |
| Occurrence of infiscentialleous relial insufficiency V2; ff (%) | JJ0 (J.U%) | 10/ (4.0%) | 0.0107 | 212 (3.0/0) | 220 (2.0/0) | 0.0242 | 010 (3.5%) | 413 (3.3/0) | 0.032 |

| Occurrence of chronic renal insufficiency w/o CKD (for PS) | 306 (4.6%) | 164 (4.0%) | 0.0296 | 201 (2.2%) | 164 (1.9%) | 0.0212 | 507 (3.2%) | 328 (2.6%) | 0.036 |
|---|---|---|---|---|---|---|---|---|---|
| Chronic kidney disease Stage 1-2 (for PS); n (%) | 176 (2.6%) | 62 (1.5%) | 0.0777 | 78 (0.9%) | 65 (0.8%) | 0.0109 | 254 (1.6%) | 127 (1.0%) | 0.053 |
| CKD stage 3-6 + dialysis (for PS); n (%) | 443 (6.6%) | 146 (3.6%) | 0.1367 | 256 (2.8%) | 168 (2.0%) | 0.0523 | 699 (4.4%) | 314 (2.5%) | 0.104 |
| Bladder stones+Kidney stones (for PS); n (%) | 133 (2.0%) | 76 (1.9%) | 0.0072 | 155 (1.7%) | 155 (1.8%) | -0.0076 | 288 (1.8%) | 231 (1.8%) | 0.000 |
| Urinary tract infections (UTIs); n (%) | 322 (4.8%) | 151 (3.7%) | 0.0545 | 256 (2.8%) | 265 (3.1%) | -0.0177 | 578 (3.7%) | 416 (3.3%) | 0.022 |
| Edema; n (%) | 230 (3.4%) | 110 (2.7%) | 0.0407 | 202 (2.2%) | 159 (1.9%) | 0.0212 | 432 (2.7%) | 269 (2.1%) | 0.039 |
| Other comorbidities | | | | <u> </u> | | | | | |
| COPD; n (%) | 860 (12.8%) | 431 (10.6%) | 0.0685 | 643 (7.1%) | 560 (6.5%) | 0.0238 | 1,503 (9.5%) | 991 (7.8%) | 0.061 |
| Asthma; n (%) | 438 (6.5%) | 253 (6.2%) | 0.0123 | 445 (4.9%) | 371 (4.3%) | 0.0286 | 883 (5.6%) | 624 (4.9%) | 0.031 |
| Obstructive sleep apnea; n (%) | 711 (10.6%) | 388 (9.5%) | 0.0366 | 818 (9.1%) | 674 (7.9%) | 0.0430 | 1,529 (9.7%) | 1,062 (8.4%) | 0.045 |
| Pneumonia; n (%) | 281 (4.2%) | 136 (3.3%) | 0.0474 | 244 (2.7%) | 212 (2.5%) | 0.0126 | 525 (3.3%) | 348 (2.8%) | 0.029 |
| Hyperthyroidism + Hypothyroidism + Other disorders of th | 921 (13.7%) | 441 (10.8%) | 0.0885 | 882 (9.8%) | 723 (8.4%) | 0.0487 | 1,803 (11.4%) | 1,164 (9.2%) | 0.072 |
| Liver disease; n (%) | 4 (0.1%) | 5 (0.1%) | 0.0000 | 3 (0.0%) | 1 (0.0%) | #DIV/0! | 007 (0.0%) | 006 (0.0%) | #DIV/0! |
| Osteoarthritis; n (%) | 1,078 (16.0%) | 516 (12.6%) | 0.0972 | 916 (10.1%) | 716 (8.4%) | 0.0587 | 1,994 (12.7%) | 1,232 (9.7%) | 0.095 |
| Other arthritis, arthropathies and musculoskeletal pain; n | 2,166 (32.2%) | 1,211 (29.6%) | 0.0563 | 2,538 (28.1%) | 2,206 (25.8%) | 0.0519 | 4,704 (29.9%) | 3,417 (27.0%) | 0.064 |
| Dorsopathies; n (%) | 1,508 (22.4%) | 880 (21.5%) | 0.0217 | 1,749 (19.4%) | 1,486 (17.4%) | 0.0516 | 3,257 (20.7%) | 2,366 (18.7%) | 0.050 |
| Fractures; n (%) | 136 (2.0%) | 68 (1.7%) | 0.0223 | 146 (1.6%) | 117 (1.4%) | 0.0165 | 282 (1.8%) | 185 (1.5%) | 0.024 |
| Falls v2; n (%) | 127 (1.9%) | 45 (1.1%) | 0.0659 | 56 (0.6%) | 35 (0.4%) | 0.0284 | 183 (1.2%) | 080 (0.6%) | 0.064 |
| Osteoporosis; n (%) | 197 (2.9%) | 80 (2.0%) | 0.0582 | 120 (1.3%) | 72 (0.8%) | 0.0491 | 317 (2.0%) | 152 (1.2%) | 0.064 |
| Depression; n (%) | 635 (9.4%) | 382 (9.4%) | 0.0000 | 575 (6.4%) | 566 (6.6%) | -0.0081 | 1,210 (7.7%) | 948 (7.5%) | 0.008 |
| Anxiety; n (%) | 875 (13.0%) | 465 (11.4%) | 0.0489 | 804 (8.9%) | 608 (7.1%) | 0.0664 | 1,679 (10.7%) | 1,073 (8.5%) | 0.075 |
| Sleep_Disorder; n (%) | 255 (3.8%) | 315 (7.7%) | -0.1681 | 477 (5.3%) | 702 (8.2%) | -0.1158 | 732 (4.6%) | 1,017 (8.0%) | -0.140 |
| Dementia; n (%) | 118 (1.8%) | 34 (0.8%) | 0.0884 | 46 (0.5%) | 31 (0.4%) | 0.0149 | 164 (1.0%) | 065 (0.5%) | 0.058 |
| Delirium; n (%) | 60 (0.9%) | 27 (0.7%) | 0.0225 | 44 (0.5%) | 33 (0.4%) | 0.0149 | 104 (0.7%) | 060 (0.5%) | 0.026 |
| Psychosis; n (%) | 37 (0.6%) | 19 (0.5%) | 0.0135 | 25 (0.3%) | 17 (0.2%) | 0.0200 | 062 (0.4%) | 036 (0.3%) | 0.017 |
| Use of medications | | | | | | | | | |
| Use of ACE inhibitors; n (%) | 3,343 (49.7%) | 2,234 (54.7%) | -0.1002 | 4,901 (54.3%) | 4,985 (58.3%) | -0.0807 | 8,244 (52.4%) | 7,219 (57.1%) | -0.095 |
| Use of ARBs; n (%) | 1,464 (21.8%) | 735 (18.0%) | 0.0953 | 1,721 (19.1%) | 1,420 (16.6%) | 0.0653 | 3,185 (20.2%) | 2,155 (17.0%) | 0.082 |
| Use of Loop Diuretics - United; n (%) | 620 (9.2%) | 250 (6.1%) | 0.1168 | 536 (5.9%) | 483 (5.6%) | 0.0129 | 1,156 (7.3%) | 733 (5.8%) | 0.061 |
| Use of other diuretics- United; n (%) | 273 (4.1%) | 151 (3.7%) | 0.0207 | 348 (3.9%) | 318 (3.7%) | 0.0105 | 621 (3.9%) | 469 (3.7%) | 0.010 |
| Use of nitrates-United; n (%) | 2,800 (41.7%) | 1,806 (44.2%) | -0.0505 | 3,934 (43.6%) | 3,837 (44.8%) | -0.0242 | 6,734 (42.8%) | 5,643 (44.6%) | -0.036 |
| Use of other hypertension drugs; n (%) | 295 (4.4%) | 145 (3.5%) | 0.0462 | 292 (3.2%) | 293 (3.4%) | -0.0112 | 587 (3.7%) | 438 (3.5%) | 0.011 |
| Use of digoxin- United; n (%) | 52 (0.8%) | 34 (0.8%) | 0.0000 | 40 (0.4%) | 49 (0.6%) | -0.0284 | 092 (0.6%) | 083 (0.7%) | -0.012 |
| Use of Anti-arrhythmics; n (%) | 144 (2.1%) | 71 (1.7%) | 0.0293 | 122 (1.4%) | 159 (1.9%) | -0.0393 | 266 (1.7%) | 230 (1.8%) | -0.008 |
| Use of COPD/asthma meds- United; n (%) | 844 (12.6%) | 485 (11.9%) | 0.0214 | 971 (10.8%) | 928 (10.8%) | 0.0000 | 1,815 (11.5%) | 1,413 (11.2%) | 0.009 |
| Use of statins; n (%) | 6,084 (90.5%) | 3,736 (91.5%) | -0.0349 | 8,217 (91.0%) | 7,798 (91.1%) | -0.0035 | 14,301 (90.8%) | 11,534 (91.2%) | -0.014 |
| Use of other lipid-lowering drugs; n (%) | 442 (6.6%) | 340 (8.3%) | -0.0648 | 695 (7.7%) | 801 (9.4%) | -0.0608 | 1,137 (7.2%) | 1,141 (9.0%) | -0.066 |
| Use of antiplatelet agents; n (%) | 532 (7.9%) | 340 (8.3%) | -0.0147 | 616 (6.8%) | 695 (8.1%) | -0.0495 | 1,148 (7.3%) | 1,035 (8.2%) | -0.034 |
| Use of oral anticoagulants (Dabigatran, Rivaroxaban, Apix | <del></del> | 81 (2.0%) | 0.0865 | 230 (2.5%) | 210 (2.5%) | 0.0000 | 460 (2.9%) | 291 (2.3%) | 0.038 |
| Use of heparin and other low-molecular weight heparins; | 27 (0.4%) | 11 (0.3%) | 0.0169 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 027 (0.2%) | 011 (0.1%) | 0.026 |
| Use of NSAIDs; n (%) | 996 (14.8%) | 539 (13.2%) | 0.0461 | 1,386 (15.4%) | 1,189 (13.9%) | 0.0424 | 2,382 (15.1%) | 1,728 (13.7%) | 0.040 |
| Use of oral corticosteroids; n (%) | 1,091 (16.2%) | 556 (13.6%) | 0.0731 | 1,337 (14.8%) | 1,173 (13.7%) | 0.0315 | 2,428 (15.4%) | 1,729 (13.7%) | 0.048 |
| Use of bisphosphonate (United); n (%) | 75 (1.1%) | 33 (0.8%) | 0.0309 | 46 (0.5%) | 42 (0.5%) | 0.0000 | 121 (0.8%) | 075 (0.6%) | 0.024 |
| Use of opioids- United; n (%) | 1,316 (19.6%) | 924 (22.6%) | -0.0736 | 1,852 (20.5%) | 1,859 (21.7%) | -0.0294 | 3,168 (20.1%) | 2,783 (22.0%) | -0.047 |
| Use of antidepressants; n (%) | 1,106 (16.5%) | 650 (15.9%) | 0.0163 | 1,388 (15.4%) | 1,229 (14.4%) | 0.0281 | 2,494 (15.8%) | 1,879 (14.9%) | 0.025 |
| Use of antipsychotics; n (%) | 93 (1.4%) | 36 (0.9%) | 0.0469 | 86 (1.0%) | 65 (0.8%) | 0.0212 | 179 (1.1%) | 101 (0.8%) | 0.031 |
| Use of anticonvulsants; n (%) | 635 (9.4%) | 293 (7.2%) | 0.0798 | 589 (6.5%) | 494 (5.8%) | 0.0291 | 1,224 (7.8%) | 787 (6.2%) | 0.063 |
| Use of Benzos- United; n (%) | 608 (9.0%) | 383 (9.4%) | -0.0138 | 881 (9.8%) | 790 (9.2%) | 0.0205 | 1,489 (9.5%) | 1,173 (9.3%) | 0.007 |
| Use of anxiolytics/hypnotics- United; n (%) | 285 (4.2%) | 226 (5.5%) | -0.0605 | 443 (4.9%) | 467 (5.5%) | -0.0270 | 728 (4.6%) | 693 (5.5%) | -0.041 |
| Use of dementia meds- United; n (%) | 44 (0.7%) | 19 (0.5%) | 0.0259 | 27 (0.3%) | 8 (0.1%) | 0.0448 | 071 (0.5%) | 027 (0.2%) | 0.051 |

| Use of antiparkinsonian meds- United; n (%) | 118 (1.8%) | 46 (1.1%) | 0.0586 | 101 (1.1%) | 71 (0.8%) | 0.0309 | 219 (1.4%) | 117 (0.9%) | 0.047 |
|---|---|---|---|---|---|---|---|---|---|
| Use of glucose test strips; n (%) | 86 (1.3%) | 48 (1.2%) | 0.0090 | 116 (1.3%) | 113 (1.3%) | 0.0000 | 202 (1.3%) | 161 (1.3%) | 0.000 |
| Use of thiazide- United; n (%) | 537 (8.0%) | 288 (7.1%) | 0.0341 | 606 (6.7%) | 544 (6.4%) | 0.0121 | 1,143 (7.3%) | 832 (6.6%) | 0.028 |
| Use of beta blockers; n (%) | 5,753 (85.6%) | 3,550 (86.9%) | -0.0378 | 7,873 (87.2%) | 7,618 (89.0%) | -0.0556 | 13,626 (86.5%) | 11,168 (88.3%) | -0.054 |
| Use of calcium channel blockers; n (%) | 1,357 (20.2%) | 706 (17.3%) | 0.0744 | 1,642 (18.2%) | 1,370 (16.0%) | 0.0585 | 2,999 (19.0%) | 2,076 (16.4%) | 0.068 |
| Use of aspirin; n (%) | 1,042 (15.5%) | 369 (9.0%) | 0.1992 | 1,807 (20.0%) | 925 (10.8%) | 0.2570 | 2,849 (18.1%) | 1,294 (10.2%) | 0.228 |
| Use of Low Intensity Statins; n (%) | 1,500 (22.3%) | 1,250 (30.6%) | -0.1890 | 2,143 (23.7%) | 2,734 (32.0%) | -0.1860 | 3,643 (23.1%) | 3,984 (31.5%) | -0.189 |
| Use of High Intensity Statins; n (%) | 5,326 (79.2%) | 2,878 (70.5%) | 0.2015 | 7,021 (77.8%) | 5,772 (67.5%) | 0.2326 | 12,347 (78.4%) | 8,650 (68.4%) | 0.228 |
| Use of Sympatomimetic agents; n (%) | 66 (1.0%) | 45 (1.1%) | -0.0098 | 121 (1.3%) | 85 (1.0%) | 0.0281 | 187 (1.2%) | 130 (1.0%) | 0.019 |
| Use of CNS stimulants; n (%) | 27 (0.4%) | 13 (0.3%) | 0.0169 | 44 (0.5%) | 54 (0.6%) | -0.0135 | 071 (0.5%) | 067 (0.5%) | 0.000 |
| All antidiabetic medications except Insulin; n (%) | 1,603 (23.8%) | 915 (22.4%) | 0.0332 | 2,040 (22.6%) | 1,948 (22.8%) | -0.0048 | 3,643 (23.1%) | 2,863 (22.6%) | 0.012 |
| DM Medications - Insulin Copy; n (%) | 616 (9.2%) | 352 (8.6%) | 0.0211 | 817 (9.1%) | 765 (8.9%) | 0.0070 | 1,433 (9.1%) | 1,117 (8.8%) | 0.011 |
| Use of estrogens, progestins, androgens; n (%) | 195 (2.9%) | 153 (3.7%) | -0.0448 | 381 (4.2%) | 381 (4.5%) | -0.0147 | 576 (3.7%) | 534 (4.2%) | -0.026 |
| Use of Angiogenesis inhibitors; n (%) | 4 (0.1%) | 0 (0.0%) | 0.0447 | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 005 (0.0%) | 000 (0.0%) | #DIV/0! |
| | 7 (0.1%) | 4 (0.1%) | 0.0000 | 18 (0.2%) | 15 (0.2%) | 0.0000 | 025 (0.2%) | 019 (0.2%) | 0.000 |
| Use of Oral Immunosuppressants; n (%) Use of fondaparinux or Bivalirudin; n (%) | 0 (0.0%) | 2 (0.0%) | #DIV/0! | 0 (0.0%) | 2 (0.0%) | #DIV/0! | 000 (0.0%) | 004 (0.0%) | #DIV/0! |
| Use of other direct thrombin inhibitors (lepirudin, desirudi | ` ' | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| \ | ` ' | · , | 0.0000 | 1,373 (15.2%) | ` ' | 0.0028 | 2,436 (15.5%) | 1,940 (15.3%) | 0.006 |
| Use of CYP inhibitors; n (%) | 1,063 (15.8%) | 645 (15.8%) | | , , , | 1,295 (15.1%) | | | | -0.017 |
| Use of CYP inducers; n (%) | 19 (0.3%) | 14 (0.3%) | 0.0000 | 27 (0.3%) | 33 (0.4%) | -0.0169 | 046 (0.3%) | 047 (0.4%) | -0.017 |
| Burden of disease/Healthcare utilization Combined comorbidity score, 180 days Copy | | | | | | | | | |
| , | 1 F1 /1 OC) | 0.02 (1.74) | 0.3130 | 0.74 (1.54) | 0.50 (1.42) | 0.1615 | 1.07 (1.73) | 0.64 (1.54) | 0.263 |
| mean (sd) | 1.51 (1.96) | 0.93 (1.74) | 0.0000 | 0.74 (1.54) | 0.50 (1.43) | 0.0000 | 0.43 (1.73) | 0.32 (1.54) | 0.263 |
| median [IQR] | 1.00 [0.00, 3.00] | 1.00 [0.00, 2.00] | 0.0000 | 0.00 [0.00, 2.00] | 0.00 [-1.00, 1.00] | 0.0000 | 0.45 (1.75) | 0.32 (1.34) | 0.067 |
| Frailty Score (mean): Empirical Version 365 days, v2 | 0.10 (0.04) | 0.17 (0.04) | 0.3500 | 0.17 (0.03) | 0.17 (0.03) | 0.0000 | 0.17 (0.03) | 0.17 (0.03) | 0.000 |
| mean (sd) | 0.18 (0.04) | 0.17 (0.04) | 0.2500 | 0.17 (0.03) | 0.17 (0.03) | | | | 0.000 |
| median [IQR] | 0.17 [0.15, 0.20] | 0.17 [0.15, 0.19] | 0.0000 | 0.16 [0.15, 0.19] | 0.16 [0.14, 0.18] | 0.0000 | 0.16 (0.03) | 0.16 (0.03) | 0.000 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd digit level | | C 44 (0 40) | 0.5343 | 7.66 (0.06) | 4.42.(7.00) | 0.4268 | 9.09 (8.48) | 5.06 (7.46) | 0.505 |
| mean (sd) | 11.01 (9.01) | 6.41 (8.19) | | 7.66 (8.06) | 4.42 (7.09) | 0.4268 | | | 0.844 |
| median [IQR] | 10.00 [4.00, 17.00] | 3.00 [0.00, 11.00] | 0.8130 | 6.00 [0.00, 14.00] | 0.00 [0.00, 9.00] | 0.7905 | 7.71 (8.48) | 0.97 (7.46) | 0.844 |
| HAS-BLED Score (ICD-9 and ICD-10), 180 days | 2 50 (0 50) | 2 25 (0 56) | 0.2631 | 2.40 (0.40) | 2.4.4 (0.4.4) | 0.0869 | 3.32 (0.53) | 3.21 (0.48) | 0.218 |
| mean (sd) | 3.50 (0.58) | 3.35 (0.56) | | 3.18 (0.48) | 3.14 (0.44) | | | | 0.000 |
| median [IQR] | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.0000 | 3.00 [3.00, 3.00] | 3.00 [3.00, 3.00] | 0.0000 | 3.00 (0.53) | 3.00 (0.48) | 0.000 |
| number of different/distinct medication prescriptions | 0.04 (4.40) | 0.52 (4.22) | 0.0931 | 0.71 (4.21) | 0.50 (4.10) | 0.0405 | 0.01 (4.20) | 0 [1 (4 22) | 0.070 |
| mean (sd) | 8.94 (4.49) | 8.53 (4.32) | | 8.71 (4.31) | 8.50 (4.18) | 0.0495<br>0.0000 | 8.81 (4.39)<br>8.00 (4.39) | 8.51 (4.23) | 0.000 |
| median [IQR] | 8.00 [6.00, 11.00] | 8.00 [5.00, 11.00] | 0.0000 | 8.00 [6.00, 11.00] | 8.00 [5.00, 11.00] | | ` ' | 8.00 (4.23) | |
| Any hospitalization within prior 30 days; n (%) | 6,722 (100.0%) | 4,085 (100.0%) | #DIV/0! | 9,025 (100.0%) | 8,557 (100.0%) | #DIV/0! | 15,747 (100.0%) | 12,642 (100.0%) | #DIV/0! |
| Number of Hospitalizations | 1.00 (0.00) | 1.00 (0.00) | 0.0000 | 1.05 (0.05) | 1.00 (0.00) | 0.0726 | 1.07.(0.30) | 1.00 (0.30) | -0.034 |
| mean (sd) | 1.08 (0.30) | 1.08 (0.32) | 0.0000 | 1.06 (0.26) | 1.08 (0.29) | -0.0726 | 1.07 (0.28) | 1.08 (0.30)<br>1.00 (0.30) | 0.000 |
| median [IQR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.0000 | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.0000 | 1.00 (0.28) | 1.00 (0.30) | 0.000 |
| Number of hospital days | 2.60 (4.04) | 2 64 (4 04) | 0.0053 | 2.42.(4.04) | 2 60 (4 00) | 0.0000 | 2.50 (4.00) | 2.00 (4.05) | 0.054 |
| mean (sd) | 3.60 (1.94) | 3.61 (1.94) | -0.0052 | 3.42 (1.84) | 3.60 (1.80) | -0.0989 | 3.50 (1.88) | 3.60 (1.85) | -0.054<br>0.000 |
| median [IQR] | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.0000 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.0000 | 3.00 (1.88) | 3.00 (1.85) | 0.000 |
| Number of Emergency Department (ED) visits v3 | 1.07 (1.20) | 1.05 (1.00) | 0.0076 | 2.52.(5.62) | 2 24 (5 25) | 0.0250 | 2.47.(4.25) | 2.50 (5.02) | -0.023 |
| mean (sd) | 1.07 (1.30) | 1.06 (1.32) | 0.0076 | 3.52 (5.63) | 3.31 (6.05) | 0.0359 | 2.47 (4.35) | 2.58 (5.03) | -0.023 |
| median [IQR] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.0000 | 2.00 [0.00, 4.00] | 2.00 [0.00, 4.00] | 0.0000 | 1.57 (4.35) | 1.68 (5.03) | -0.023 |
| Number of Office visits | 2.42./2.46 | 2.02.(2.22) | 0.0010 | 2.77 (2.04) | 2.67.(2.02) | 0.0344 | 2.02.(2.04) | 2.75 (2.00) | 0.050 |
| mean (sd) | 3.12 (3.16) | 2.92 (3.33) | 0.0616 | 2.77 (2.94) | 2.67 (2.93) | 0.0341 | 2.92 (3.04) | 2.75 (3.06) | 0.056 |
| median [IQR] | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 0.0000 | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 0.0000 | 2.00 (3.04) | 2.00 (3.06) | 0.000 |
| Number of internal medicine/family medicine visits | 7.44 (40.6%) | 5 72 (2.66) | 0.4272 | 2.02 (5.05) | 2.75 (0.66) | 0.0000 | F 20 (2.44) | 4 20 (7 70) | 0.413 |
| mean (sd) | 7.11 (10.84) | 5.72 (9.60) | 0.1358 | 3.93 (5.98) | 3.75 (6.60) | 0.0286 | 5.29 (8.41) | 4.39 (7.70) | 0.112 |
| median [IQR] | 4.00 [1.00, 9.00] | 3.00 [0.00, 7.00] | 0.0977 | 2.00 [0.00, 5.00] | 2.00 [0.00, 5.00] | 0.0000 | 2.85 (8.41) | 2.32 (7.70) | 0.066 |

| Number of Cardiologist visits | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | 8.41 (5.38) | 8.07 (4.88) | 0.0662 | 1.06 (2.17) | 0.97 (2.18) | 0.0414 | 4.20 (3.88) | 3.26 (3.30) | 0.261 |
| median [IQR] | 8.00 [5.00, 11.00] | 7.00 [5.00, 10.00] | 0.1947 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.0000 | 3.41 (3.88) | 2.26 (3.30) | 0.319 |
| Number electrocardiograms received v2 | 0.00 [5.00, 11.00] | 7.00 [5.00, 10.00] | | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | | 0112 (0100) | ==== (====) | |
| mean (sd) | 3.28 (2.45) | 3.32 (2.52) | -0.0161 | 0.98 (1.33) | 1.05 (1.40) | -0.0513 | 1.96 (1.89) | 1.78 (1.84) | 0.097 |
| median [IQR] | 3.00 [2.00, 4.00] | 3.00 [2.00, 5.00] | 0.0000 | 1.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | 0.0000 | 1.85 (1.89) | 1.65 (1.84) | 0.107 |
| Number of BNP tests | | | | | | | ` , | , , | |
| mean (sd) | 0.10 (0.37) | 0.10 (0.37) | 0.0000 | 0.12 (0.38) | 0.13 (0.39) | -0.0260 | 0.11 (0.38) | 0.12 (0.38) | -0.026 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.38) | 0.00 (0.38) | 0.000 |
| Number of Cardiac biomarkers tests (tropnin, CK-MBs, My | | | | | . , , | | | | |
| mean (sd) | 0.68 (1.66) | 0.76 (1.77) | -0.0466 | 0.69 (1.61) | 0.83 (1.79) | -0.0822 | 0.69 (1.63) | 0.81 (1.78) | -0.070 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.00 (1.63) | 0.00 (1.78) | 0.000 |
| Number of Ambulatory Blood pressure monitoring tests | | | | | . , , | | | | |
| mean (sd) | 0.00 (0.02) | 0.00 (0.02) | 0.0000 | 0.00 (0.04) | 0.00 (0.03) | 0.0000 | 0.00 (0.03) | 0.00 (0.03) | 0.000 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.03) | 0.00 (0.03) | 0.000 |
| N of days on antihypertensive medications during baseling | | | | | | | | | |
| mean (sd) | 81.19 (79.68) | 71.98 (77.47) | 0.1172 | 74.18 (78.62) | 68.85 (77.22) | 0.0684 | 77.17 (79.07) | 69.86 (77.30) | 0.093 |
| median [IQR] | 62.50 [1.00, 172.00] | 21.00 [1.00, 164.00] | 0.5281 | 29.00 [1.00, 167.00] | 8.00 [1.00, 162.00] | 0.2695 | 43.30 (79.07) | 12.20 (77.30) | 0.398 |
| N of days in database anytime prior | | | | | | | | | |
| mean (sd) | 1,685.49 (1,370.91) | 1,619.30 (1,246.27) | 0.0505 | 2,118.05 (1,473.24) | 1,786.28 (1,260.85) | 0.2420 | 1933.40 (1430.45) | 1732.32 (1256.16) | 0.149 |
| median [IQR] | 1,246.00 [606.00, 2, | 41,242.00 [605.00, 2,4 | 0.0031 | 1,804.00 [830.00, 3,2 | 1,443.00 [726.00, 2,7 | 0.2633 | 1565.80 (1430.45) | 1378.05 (1256.16) | 0.139 |
| Mean Copay for per prescription cost (charges in U.S. \$) ( | 1 | | | | | | | | |
| mean (sd) | 21.80 (31.56) | 25.04 (28.00) | -0.1086 | 15.43 (20.81) | 18.99 (25.39) | -0.1534 | 18.15 (25.95) | 20.94 (26.26) | -0.107 |
| median [IQR] | 13.33 [5.00, 27.78] | 17.11 [7.40, 33.33] | -0.1267 | 10.00 [1.98, 21.01] | 12.44 [4.50, 25.29] | -0.1051 | 11.42 (25.95) | 13.95 (26.26) | -0.097 |
| Missing; n (%) | 879 (13.1%) | 638 (15.6%) | -0.0714 | 1,391 (15.4%) | 1,411 (16.5%) | -0.0300 | 2,270 (14.4%) | 2,049 (16.2%) | -0.050 |
| Duration of index hospitalization (i.e. anchor hospitalizati | | , , | | | , , | | | | |
| mean (sd) | 1.00 (0.00) | 1.00 (0.00) | #DIV/0! | 1.00 (0.00) | 1.00 (0.00) | #DIV/0! | 1.00 (0.00) | 1.00 (0.00) | #DIV/0! |
| median [IQR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | #DIV/0! | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | #DIV/0! | 1.00 (0.00) | 1.00 (0.00) | #DIV/0! |
| N of Generic name drugs | | | | | | | | | |
| mean (sd) | 13.03 (11.49) | 11.70 (10.59) | 0.1204 | 11.38 (9.78) | 10.30 (8.90) | 0.1155 | 12.08 (10.54) | 10.75 (9.48) | 0.133 |
| median [IQR] | 10.00 [5.00, 17.00] | 8.00 [4.00, 16.00] | 0.1810 | 9.00 [5.00, 15.00] | 8.00 [4.00, 14.00] | 0.1069 | 9.43 (10.54) | 8.00 (9.48) | 0.143 |
| N of Brand name drugs | | | | | | | | | |
| mean (sd) | 3.08 (3.59) | 3.51 (4.09) | -0.1117 | 3.42 (3.62) | 3.99 (4.24) | -0.1446 | 3.27 (3.61) | 3.83 (4.19) | -0.143 |
| median [IQR] | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 0.0000 | 2.00 [1.00, 4.00] | 2.00 [1.00, 5.00] | 0.0000 | 2.00 (3.61) | 2.00 (4.19) | 0.000 |
| Number of D-dimer tests | | | | | | | | | |
| mean (sd) | 0.06 (0.25) | 0.06 (0.25) | 0.0000 | 0.07 (0.28) | 0.07 (0.29) | 0.0000 | 0.07 (0.27) | 0.07 (0.28) | 0.000 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.27) | 0.00 (0.28) | 0.000 |
| Numbe of CRP, high-sensitivity CRP tests | | | | | | | | | |
| mean (sd) | 0.05 (0.30) | 0.04 (0.33) | 0.0317 | 0.04 (0.27) | 0.04 (0.26) | 0.0000 | 0.04 (0.28) | 0.04 (0.28) | 0.000 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.28) | 0.00 (0.28) | 0.000 |
| Number of PT or aPTTt tests | | | | | | | | | |
| mean (sd) | 0.39 (1.09) | 0.36 (0.99) | 0.0288 | 0.37 (0.92) | 0.44 (1.04) | -0.0713 | 0.38 (1.00) | 0.41 (1.02) | -0.030 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.00 (1.00) | 0.00 (1.02) | 0.000 |
| Number of Bleeding time tests | ļ | | | | | | | | |
| mean (sd) | 0.00 (0.02) | 0.00 (0.00) | 0.0000 | 0.00 (0.01) | 0.00 (0.00) | 0.0000 | 0.00 (0.02) | 0.00 (0.00) | 0.000 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.02) | 0.00 (0.00) | 0.000 |
| Occurrence of creatinine tests ordered (for PS); n (%) | 227 (3.4%) | 107 (2.6%) | 0.0469 | 228 (2.5%) | 265 (3.1%) | -0.0364 | 455 (2.9%) | 372 (2.9%) | 0.000 |
| Cardiovascular stress test; n (%) | 15 (0.2%) | 6 (0.1%) | 0.0258 | 15 (0.2%) | 15 (0.2%) | 0.0000 | 030 (0.2%) | 021 (0.2%) | 0.000 |
| Echocardiogram; n (%) | 5,099 (75.9%) | 2,718 (66.5%) | 0.2087 | 6,478 (71.8%) | 5,447 (63.7%) | 0.1739 | 11,577 (73.5%) | 8,165 (64.6%) | 0.193 |
| Colonoscopy; n (%) | 222 (3.3%) | 152 (3.7%) | -0.0218 | 329 (3.6%) | 294 (3.4%) | 0.0109 | 551 (3.5%) | 446 (3.5%) | 0.000 |
| Fecal occult blood (FOB) test; n (%) | 163 (2.4%) | 115 (2.8%) | -0.0251 | 224 (2.5%) | 226 (2.6%) | -0.0063 | 387 (2.5%) | 341 (2.7%) | -0.013 |

| Flu vaccine; n (%) | 978 (14.5%) | 523 (12.8%) | 0.0495 | 768 (8.5%) | 687 (8.0%) | 0.0182 | 1,746 (11.1%) | 1,210 (9.6%) | 0.049 |
|---|---|---|---|---|---|---|---|---|---|
| Mammogram; n (%) | 396 (5.9%) | 170 (4.2%) | 0.0777 | 369 (4.1%) | 301 (3.5%) | 0.0314 | 765 (4.9%) | 471 (3.7%) | 0.059 |
| Pap smear; n (%) | 132 (2.0%) | 85 (2.1%) | -0.0071 | 174 (1.9%) | 182 (2.1%) | -0.0143 | 306 (1.9%) | 267 (2.1%) | -0.014 |
| Pneumonia vaccine; n (%) | 1,315 (19.6%) | 496 (12.1%) | 0.2065 | 754 (8.4%) | 461 (5.4%) | 0.1186 | 2,069 (13.1%) | 957 (7.6%) | 0.181 |
| PSA test or Prostate exam for DRE; n (%) | 1,018 (15.1%) | 646 (15.8%) | -0.0194 | 1,125 (12.5%) | 1,167 (13.6%) | -0.0327 | 2,143 (13.6%) | 1,813 (14.3%) | -0.020 |
| Bone mineral density; n (%) | 110 (1.6%) | 60 (1.5%) | 0.0081 | 79 (0.9%) | 47 (0.5%) | 0.0480 | 189 (1.2%) | 107 (0.8%) | 0.040 |
| Drug eluting stent; n (%) | 998 (14.8%) | 1,987 (48.6%) | -0.7796 | 2,503 (27.7%) | 3,877 (45.3%) | -0.3718 | 3,501 (22.2%) | 5,864 (46.4%) | -0.527 |
| Bare metal stent; n (%) | 5,844 (86.9%) | 2,853 (69.8%) | 0.4244 | 7,737 (85.7%) | 4,842 (56.6%) | 0.6782 | 13,581 (86.2%) | 7,695 (60.9%) | 0.599 |

| | | Optum | | | Marketscan | | | Pooled | |
|---|---|---|---|---|---|---|---|---|---|
| | Ticagrelor | Prasugrel | St. Diff | Ticagrelor | Prasugrel | St. Diff | Ticagrelor | Prasugrel | St. Diff |
| Number of patients | 2,498 | 2,498 | | 4,802 | 4,802 | | 7,300 | 7,300 | |
| Quarter/Year of Cohort Entry Date | | | | | | | | | |
| Q3 2011; n (%) | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 2 (0.0%) | 2 (0.0%) | #DIV/0! | 003 (0.0%) | 002 (0.0%) | #DIV/0! |
| Q4 2011; n (%) | 2 (0.1%) | 2 (0.1%) | 0.0000 | 19 (0.4%) | 20 (0.4%) | 0.0000 | 021 (0.3%) | 022 (0.3%) | 0.000 |
| Q1 2012; n (%) | 11 (0.4%) | 16 (0.6%) | -0.0284 | 51 (1.1%) | 42 (0.9%) | 0.0201 | 062 (0.8%) | 058 (0.8%) | 0.000 |
| Q2 2012; n (%) | 30 (1.2%) | 23 (0.9%) | 0.0294 | 104 (2.2%) | 98 (2.0%) | 0.0139 | 134 (1.8%) | 121 (1.7%) | 0.008 |
| Q3 2012; n (%) | 44 (1.8%) | 51 (2.0%) | -0.0146 | 142 (3.0%) | 156 (3.2%) | -0.0115 | 186 (2.5%) | 207 (2.8%) | -0.019 |
| Q4 2012; n (%) | 42 (1.7%) | 54 (2.2%) | -0.0362 | 177 (3.7%) | 189 (3.9%) | -0.0105 | 219 (3.0%) | 243 (3.3%) | -0.017 |
| Q1 2013; n (%) | 78 (3.1%) | 67 (2.7%) | 0.0238 | 171 (3.6%) | 176 (3.7%) | -0.0053 | 249 (3.4%) | 243 (3.3%) | 0.006 |
| Q2 2013; n (%) | 89 (3.6%) | 78 (3.1%) | 0.0278 | 188 (3.9%) | 190 (4.0%) | -0.0051 | 277 (3.8%) | 268 (3.7%) | 0.005 |
| Q3 2013; n (%) | 70 (2.8%) | 71 (2.8%) | 0.0000 | 243 (5.1%) | 253 (5.3%) | -0.0090 | 313 (4.3%) | 324 (4.4%) | -0.005 |
| Q4 2013; n (%) | 75 (3.0%) | 73 (2.9%) | 0.0059 | 249 (5.2%) | 235 (4.9%) | 0.0137 | 324 (4.4%) | 308 (4.2%) | 0.010 |
| Q1 2014; n (%) | 77 (3.1%) | 74 (3.0%) | 0.0058 | 224 (4.7%) | 223 (4.6%) | 0.0047 | 301 (4.1%) | 297 (4.1%) | 0.000 |
| Q2 2014; n (%) | 79 (3.2%) | 70 (2.8%) | 0.0235 | 258 (5.4%) | 265 (5.5%) | -0.0044 | 337 (4.6%) | 335 (4.6%) | 0.000 |
| Q3 2014; n (%) | 89 (3.6%) | 76 (3.0%) | 0.0336 | 278 (5.8%) | 291 (6.1%) | -0.0127 | 367 (5.0%) | 367 (5.0%) | 0.000 |
| Q4 2014; n (%) | 90 (3.6%) | 78 (3.1%) | 0.0278 | 302 (6.3%) | 285 (5.9%) | 0.0167 | 392 (5.4%) | 363 (5.0%) | 0.018 |
| Q1 2015; n (%) | 67 (2.7%) | 71 (2.8%) | -0.0061 | 186 (3.9%) | 188 (3.9%) | 0.0000 | 253 (3.5%) | 259 (3.5%) | 0.000 |
| Q2 2015; n (%) | 63 (2.5%) | 62 (2.5%) | 0.0000 | 158 (3.3%) | 166 (3.5%) | -0.0110 | 221 (3.0%) | 228 (3.1%) | -0.006 |
| Q3 2015; n (%) | 78 (3.1%) | 77 (3.1%) | 0.0000 | 205 (4.3%) | 191 (4.0%) | 0.0150 | 283 (3.9%) | 268 (3.7%) | 0.010 |
| Q4 2015; n (%) | 100 (4.0%) | 90 (3.6%) | 0.0209 | 249 (5.2%) | 234 (4.9%) | 0.0137 | 349 (4.8%) | 324 (4.4%) | 0.019 |
| Q1 2016; n (%) | 84 (3.4%) | 91 (3.6%) | -0.0109 | 263 (5.5%) | 244 (5.1%) | 0.0179 | 347 (4.8%) | 335 (4.6%) | 0.009 |
| Q2 2016; n (%) | 97 (3.9%) | 102 (4.1%) | -0.0102 | 236 (4.9%) | 230 (4.8%) | 0.0047 | 333 (4.6%) | 332 (4.5%) | 0.005 |
| Q3 2016; n (%) | 104 (4.2%) | 112 (4.5%) | -0.0147 | 249 (5.2%) | 232 (4.8%) | 0.0184 | 353 (4.8%) | 344 (4.7%) | 0.005 |
| Q4 2016; n (%) | 129 (5.2%) | 123 (4.9%) | 0.0137 | 216 (4.5%) | 225 (4.7%) | -0.0095 | 345 (4.7%) | 348 (4.8%) | -0.005 |
| Q1 2017; n (%) | 100 (4.0%) | 113 (4.5%) | -0.0248 | 141 (2.9%) | 158 (3.3%) | -0.0231 | 241 (3.3%) | 271 (3.7%) | -0.022 |
| Q2 2017; n (%) | 110 (4.4%) | 122 (4.9%) | -0.0237 | 159 (3.3%) | 162 (3.4%) | -0.0056 | 269 (3.7%) | 284 (3.9%) | -0.010 |
| Q3 2017; n (%) | 119 (4.8%) | 125 (5.0%) | -0.0093 | 173 (3.6%) | 192 (4.0%) | -0.0209 | 292 (4.0%) | 317 (4.3%) | -0.015 |
| | 107 (4.3%) | 122 (4.9%) | -0.0286 | 158 (3.3%) | 154 (3.2%) | 0.0056 | 265 (3.6%) | 276 (3.8%) | -0.013 |
| Q4 2017; n (%)<br>Q1 2018; n (%) | 92 (3.7%) | 96 (3.8%) | -0.0280 | 1 (0.0%) | 1 (0.0%) | #DIV/0! | 093 (1.3%) | 097 (1.3%) | 0.000 |
| | 92 (3.7%) | 90 (3.6%) | -0.0055 | 1 (0.0%) | 1 (0.0%) | #DIV/U! | 093 (1.3%) | 097 (1.370) | 0.000 |
| Demographics Age | | | | | | | | | |
| mean (sd) | 61.84 (11.27) | 61.48 (10.03) | 0.0337 | 57.39 (9.86) | 57.47 (8.66) | -0.0086 | 58.91 (10.36) | 58.84 (9.15) | 0.007 |
| median [IQR] | · | 62.00 [55.00, 69.00] | 0.0000 | 58.00 [51.00, 63.00] | , , | 0.0000 | 59.37 (10.36) | 59.37 (9.15) | 0.000 |
| Gender without zero category- United | 02.00 [54.00, 70.00] | 02.00 [33.00, 03.00] | 0.0000 | 30.00 [31.00, 03.00] | 30.00 [32.00, 03.00] | 0.0000 | 33.37 (20.33) | 33.37 (3.23) | 0.000 |
| Males; n (%) | 1,877 (75.1%) | 1,880 (75.3%) | -0.0046 | 3,759 (78.3%) | 3,743 (77.9%) | 0.0005 | 5,636 (77.2%) | 5,623 (77.0%) | 0.005 |
| Females; n (%) | 621 (24.9%) | 618 (24.7%) | 0.0046 | 1,043 (21.7%) | 1,059 (22.1%) | 0.0005 | 1,664 (22.8%) | 1,677 (23.0%) | -0.005 |
| Region without zero category- United v3 (lumping missing | | 010 (24.770) | 0.00.0 | 1,043 (21.770) | 1,033 (22.170) | 0.0000 | 2,001 (22.070) | 2,077 (201070) | 0.005 |
| Northeast; n (%) | 234 (9.4%) | 215 (8.6%) | 0.0280 | 784 (16.3%) | 779 (16.2%) | 0.0027 | 1,018 (13.9%) | 994 (13.6%) | 0.009 |
| South; n (%) | 1,185 (47.4%) | 1,187 (47.5%) | -0.0020 | 2,159 (45.0%) | 2,186 (45.5%) | -0.0100 | 3,344 (45.8%) | 3,373 (46.2%) | -0.008 |
| Midwest; n (%) | 576 (23.1%) | 584 (23.4%) | -0.0071 | 1,178 (24.5%) | 1,165 (24.3%) | 0.0047 | 1,754 (24.0%) | 1,749 (24.0%) | 0.000 |
| West; n (%) | 503 (20.1%) | 512 (20.5%) | -0.0099 | 629 (13.1%) | 614 (12.8%) | 0.0089 | 1,132 (15.5%) | 1,126 (15.4%) | 0.003 |
| Metropolitan Statistical Area - Urban (any MSA) vs Rural | ` ' | - (/-) | | (/-) | . (==:=/=/ | | , , , | , , , , , , | |
| Urban; n (%) | 1 | | | 3,606 (75.1%) | 3,607 (75.1%) | 0.0000 | 3,606 (75.1%) | 3,607 (75.1%) | 0.0000 |
| Rural; n (%) | | | | 204 (4.2%) | 207 (4.3%) | -0.0050 | 204 (4.2%) | 207 (4.3%) | -0.0050 |
| Unknown/Missing; n (%) | | | | 992 (20.7%) | 988 (20.6%) | 0.0025 | 992 (20.7%) | 988 (20.6%) | 0.0025 |
| Commercial vs Medicare Advantage- Business Type Code | | | | · | | | · | | |
| COM = COMMERCIAL; n (%) | 1,370 (54.8%) | 1,414 (56.6%) | -0.0362 | | | | 1,370 (54.8%) | 1,414 (56.6%) | -0.0362 |
| MCR = MEDICARE; n (%) | 1,128 (45.2%) | 1,084 (43.4%) | 0.0362 | | | | 1,128 (45.2%) | 1,084 (43.4%) | 0.0362 |
| MCD = MEDICAID; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | | | | 0 (0.0%) | 0 (0.0%) | #DIV/0! |

| NONE = NO BUSINESS LINE CODE (added in 2015); n (9 | %) 0 (0.0%) | 0 (0.0%) | #DIV/0! | | | | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
|---|---|---|---|---|---|---|---|---|---|
| UNK = UNKNOWN (added in 2015); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | | | | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Commercial vs Medicare Advantage- Data Type | | , , | | | | | | | |
| 1 - Fee For Service; n (%) | | | | 3,556 (74.1%) | 3,566 (74.3%) | -0.0046 | 3,556 (74.1%) | 3,566 (74.3%) | -0.0046 |
| 2 - Encounter; n (%) | | | | 419 (8.7%) | 418 (8.7%) | 0.0000 | 419 (8.7%) | 418 (8.7%) | 0.0000 |
| 3 - Medicare; n (%) | | | | 725 (15.1%) | 714 (14.9%) | 0.0056 | 725 (15.1%) | 714 (14.9%) | 0.0056 |
| 4 - Medicare Encounter; n (%) | | | | 102 (2.1%) | 104 (2.2%) | -0.0069 | 102 (2.1%) | 104 (2.2%) | -0.0069 |
| Lifestyle factors | | | | | | | | | |
| Obesity; n (%) | 647 (25.9%) | 658 (26.3%) | -0.0091 | 966 (20.1%) | 937 (19.5%) | 0.0151 | 1,613 (22.1%) | 1,595 (21.8%) | 0.007 |
| Overweight; n (%) | 134 (5.4%) | 155 (6.2%) | -0.0342 | 111 (2.3%) | 119 (2.5%) | -0.0131 | 245 (3.4%) | 274 (3.8%) | -0.021 |
| Smoking; n (%) | 1,220 (48.8%) | 1,220 (48.8%) | 0.0000 | 1,586 (33.0%) | 1,579 (32.9%) | 0.0021 | 2,806 (38.4%) | 2,799 (38.3%) | 0.002 |
| Alcohol abuse or dependence+Drug abuse or dependence | e ( 133 (5.3%) | 120 (4.8%) | 0.0228 | 157 (3.3%) | 150 (3.1%) | 0.0114 | 290 (4.0%) | 270 (3.7%) | 0.016 |
| Diabetes-related conditions | | | | | | | | | |
| Diabetic retinopathy; n (%) | 39 (1.6%) | 38 (1.5%) | 0.0081 | 61 (1.3%) | 56 (1.2%) | 0.0090 | 100 (1.4%) | 094 (1.3%) | 0.009 |
| Occurrence of Diabetic Neuropathy v2 Copy; n (%) | 138 (5.5%) | 141 (5.6%) | -0.0044 | 158 (3.3%) | 159 (3.3%) | 0.0000 | 296 (4.1%) | 300 (4.1%) | 0.000 |
| Occurrence of diabetic nephropathy V3 with ICD10 Copy; | | 112 (4.5%) | -0.0299 | 79 (1.6%) | 86 (1.8%) | -0.0155 | 176 (2.4%) | 198 (2.7%) | -0.019 |
| Hypoglycemia v2; n (%) | 18 (0.7%) | 15 (0.6%) | 0.0124 | 50 (1.0%) | 49 (1.0%) | 0.0000 | 068 (0.9%) | 064 (0.9%) | 0.000 |
| Hyperglycemia; n (%) | 205 (8.2%) | 199 (8.0%) | 0.0073 | 290 (6.0%) | 294 (6.1%) | -0.0042 | 495 (6.8%) | 493 (6.8%) | 0.000 |
| Disorders of fluid electrolyte and acid-base balance; n (% | · · · · · · | 310 (12.4%) | -0.0092 | 432 (9.0%) | 416 (8.7%) | 0.0106 | 734 (10.1%) | 726 (9.9%) | 0.007 |
| Hyperosmolar hyperglycemic nonketotic syndrome (HON | · | 9 (0.4%) | 0.0000 | 3 (0.1%) | 6 (0.1%) | 0.0000 | 012 (0.2%) | 015 (0.2%) | 0.000 |
| Diabetic Foot; n (%) | 24 (1.0%) | 20 (0.8%) | 0.0212 | 29 (0.6%) | 30 (0.6%) | 0.0000 | 053 (0.7%) | 050 (0.7%) | 0.000 |
| Skin infections v2; n (%) | 83 (3.3%) | 83 (3.3%) | 0.0000 | 157 (3.3%) | 151 (3.1%) | 0.0114 | 240 (3.3%) | 234 (3.2%) | 0.006 |
| Erectile dysfunction; n (%) | 80 (3.2%) | 82 (3.3%) | -0.0056 | 138 (2.9%) | 129 (2.7%) | 0.0121 | 218 (3.0%) | 211 (2.9%) | 0.006 |
| Diabetes with unspecified complication; n (%) | 60 (2.4%) | 65 (2.6%) | -0.0128 | 117 (2.4%) | 118 (2.5%) | -0.0065 | 177 (2.4%) | 183 (2.5%) | -0.006 |
| Diabetes mellitus without mention of complications; n (5) | , , | 854 (34.2%) | -0.0275 | 1,551 (32.3%) | 1,561 (32.5%) | -0.0043 | 2,372 (32.5%) | 2,415 (33.1%) | -0.013 |
| | - i | | -0.0273 | · | <u> </u> | -0.0043 | 099 (1.4%) | 112 (1.5%) | -0.013 |
| Diabetes with peripheral circulatory disorders+Gangrene | · · · · · · | 54 (2.2%) | 0.0000 | 55 (1.1%) | 58 (1.2%) | 0.0103 | 058 (0.8%) | 056 (0.8%) | 0.000 |
| Diabetes with other ophthalmic manifestations+Retinal<br>Cardiovascular-related conditions | ue 10 (0.4%) | 11 (0.4%) | 0.0000 | 48 (1.0%) | 45 (0.9%) | 0.0103 | 038 (0.8%) | 056 (0.8%) | 0.000 |
| Hypertension: 1 inpatient or 2 outpatient claims within 3 | 61 1 020 (77 2%) | 1,929 (77.2%) | 0.0000 | 3,455 (71.9%) | 3,453 (71.9%) | 0.0000 | 5,384 (73.8%) | 5,382 (73.7%) | 0.002 |
| | 109 (4.4%) | 104 (4.2%) | 0.0000 | 2,019 (42.0%) | <u> </u> | 0.0000 | 2,128 (29.2%) | 2,115 (29.0%) | 0.002 |
| Malignant hypertension; n (%) | ` ' | ` ' | 0.0099 | · | 2,011 (41.9%) | 0.0020 | 5,449 (74.6%) | 5,432 (74.4%) | 0.004 |
| Hyperlipidemia v2; n (%) | 2,030 (81.3%) | 2,020 (80.9%) | | 3,419 (71.2%) | 3,412 (71.1%) | _ | | <del></del> | -0.004 |
| Acute MI; n (%) | 2,312 (92.6%) | 2,315 (92.7%) | -0.0038 | 4,566 (95.1%) | 4,566 (95.1%) | 0.0000 | 6,878 (94.2%) | 6,881 (94.3%) | |
| ACS/unstable angina; n (%) | 1,044 (41.8%) | 1,017 (40.7%) | 0.0223 | 1,795 (37.4%) | 1,824 (38.0%) | -0.0124 | 2,839 (38.9%) | 2,841 (38.9%) | 0.000 |
| Old MI; n (%) | 351 (14.1%) | 343 (13.7%) | 0.0116 | 408 (8.5%) | 423 (8.8%) | -0.0107 | 759 (10.4%) | 766 (10.5%) | -0.003 |
| Stable angina; n (%) | 509 (20.4%) | 506 (20.3%) | 0.0025 | 716 (14.9%) | 717 (14.9%) | 0.0000 | 1,225 (16.8%) | 1,223 (16.8%) | 0.000 |
| Coronary atherosclerosis and other forms of chronic isch | | 2,407 (96.4%) | 0.0000 | 4,455 (92.8%) | 4,454 (92.8%) | 0.0000 | 6,863 (94.0%) | 6,861 (94.0%) | 0.000 |
| Ischemic stroke (w and w/o mention of cerebral infarction | · · · · · · | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| TIA; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| Late effects of cerebrovascular disease; n (%) | 5 (0.2%) | 5 (0.2%) | 0.0000 | 2 (0.0%) | 3 (0.1%) | -0.0447 | 007 (0.1%) | 008 (0.1%) | 0.000 |
| Heart failure (CHF); n (%) | 433 (17.3%) | 428 (17.1%) | 0.0053 | 642 (13.4%) | 641 (13.3%) | 0.0029 | 1,075 (14.7%) | 1,069 (14.6%) | 0.003 |
| Peripheral Vascular Disease (PVD) or PVD Surgery v2; n ( | | 117 (4.7%) | -0.0193 | 130 (2.7%) | 135 (2.8%) | -0.0061 | 238 (3.3%) | 252 (3.5%) | -0.011 |
| Atrial fibrillation; n (%) | 180 (7.2%) | 170 (6.8%) | 0.0157 | 194 (4.0%) | 210 (4.4%) | -0.0199 | 374 (5.1%) | 380 (5.2%) | -0.005 |
| Other cardiac dysrhythmia; n (%) | 799 (32.0%) | 772 (30.9%) | 0.0237 | 1,200 (25.0%) | 1,244 (25.9%) | -0.0207 | 1,999 (27.4%) | 2,016 (27.6%) | -0.004 |
| Hemorrhagic stroke+Other cerebrovascular disease+Cere | bi 12 (0.5%) | 12 (0.5%) | 0.0000 | 13 (0.3%) | 11 (0.2%) | 0.0200 | 025 (0.3%) | 023 (0.3%) | 0.000 |
| Other atherosclerosis+Cardiac conduction disorders+Other | er 883 (35.3%) | 880 (35.2%) | 0.0021 | 1,345 (28.0%) | 1,355 (28.2%) | -0.0044 | 2,228 (30.5%) | 2,235 (30.6%) | -0.002 |
| Previous cardiac procedure (CABG or PTCA or Stent) + His | sti 2,455 (98.3%) | 2,459 (98.4%) | -0.0079 | 4,491 (93.5%) | 4,482 (93.3%) | 0.0081 | 6,946 (95.2%) | 6,941 (95.1%) | 0.005 |
| Kidney-related conditions | | | | | | | | | |
| Occurrence of acute renal disease v2; n (%) | 169 (6.8%) | 179 (7.2%) | -0.0157 | 192 (4.0%) | 182 (3.8%) | 0.0103 | 361 (4.9%) | 361 (4.9%) | 0.000 |
| Occurrence of hypertensive nephropathy; n (%) | 160 (6.4%) | 166 (6.6%) | -0.0081 | 133 (2.8%) | 147 (3.1%) | -0.0177 | 293 (4.0%) | 313 (4.3%) | -0.015 |
| Occurrence of miscellaneous renal insufficiency v2; n (%) | | 127 (5.1%) | 0.0045 | 126 (2.6%) | 137 (2.9%) | -0.0183 | 257 (3.5%) | 264 (3.6%) | -0.005 |
| Occurrence of chronic renal insufficiency w/o CKD (for PS | · · · · · · | 114 (4.6%) | 0.0000 | 91 (1.9%) | 101 (2.1%) | -0.0143 | 206 (2.8%) | 215 (2.9%) | -0.006 |

| Chronic kidney disease Stage 1-2 (for PS); n (%) | 50 (2.0%) | 52 (2.1%) | -0.0071 | 43 (0.9%) | 47 (1.0%) | -0.0103 | 093 (1.3%) | 099 (1.4%) | -0.009 |
|---|---|---|---|---|---|---|---|---|---|
| CKD stage 3-6 + dialysis (for PS); n (%) | 133 (5.3%) | 123 (4.9%) | 0.0182 | 108 (2.2%) | 110 (2.3%) | -0.0067 | 241 (3.3%) | 233 (3.2%) | 0.006 |
| Bladder stones+Kidney stones (for PS); n (%) | 54 (2.2%) | 52 (2.1%) | 0.0069 | 92 (1.9%) | 87 (1.8%) | 0.0074 | 146 (2.0%) | 139 (1.9%) | 0.007 |
| Urinary tract infections (UTIs); n (%) | 104 (4.2%) | 115 (4.6%) | -0.0195 | 150 (3.1%) | 146 (3.0%) | 0.0058 | 254 (3.5%) | 261 (3.6%) | -0.005 |
| Edema; n (%) | 67 (2.7%) | 78 (3.1%) | -0.0238 | 97 (2.0%) | 98 (2.0%) | 0.0000 | 164 (2.2%) | 176 (2.4%) | -0.013 |
| Other comorbidities | | | | | | | , , , | , , , | |
| COPD; n (%) | 310 (12.4%) | 306 (12.2%) | 0.0061 | 324 (6.7%) | 336 (7.0%) | -0.0119 | 634 (8.7%) | 642 (8.8%) | -0.004 |
| Asthma; n (%) | 146 (5.8%) | 162 (6.5%) | -0.0291 | 220 (4.6%) | 215 (4.5%) | 0.0048 | 366 (5.0%) | 377 (5.2%) | -0.009 |
| Obstructive sleep apnea; n (%) | 259 (10.4%) | 259 (10.4%) | 0.0000 | 392 (8.2%) | 412 (8.6%) | -0.0144 | 651 (8.9%) | 671 (9.2%) | -0.010 |
| Pneumonia; n (%) | 87 (3.5%) | 87 (3.5%) | 0.0000 | 137 (2.9%) | 127 (2.6%) | 0.0183 | 224 (3.1%) | 214 (2.9%) | 0.012 |
| Hyperthyroidism + Hypothyroidism + Other disorders of the | ny 278 (11.1%) | 304 (12.2%) | -0.0343 | 429 (8.9%) | 452 (9.4%) | -0.0173 | 707 (9.7%) | 756 (10.4%) | -0.023 |
| Liver disease; n (%) | 3 (0.1%) | 2 (0.1%) | 0.0000 | 1 (0.0%) | 1 (0.0%) | #DIV/0! | 004 (0.1%) | 003 (0.0%) | 0.045 |
| Osteoarthritis; n (%) | 337 (13.5%) | 342 (13.7%) | -0.0058 | 423 (8.8%) | 424 (8.8%) | 0.0000 | 760 (10.4%) | 766 (10.5%) | -0.003 |
| Other arthritis, arthropathies and musculoskeletal pain; r | n (768 (30.7%) | 773 (30.9%) | -0.0043 | 1,282 (26.7%) | 1,303 (27.1%) | -0.0090 | 2,050 (28.1%) | 2,076 (28.4%) | -0.007 |
| Dorsopathies; n (%) | 534 (21.4%) | 556 (22.3%) | -0.0218 | 872 (18.2%) | 879 (18.3%) | -0.0026 | 1,406 (19.3%) | 1,435 (19.7%) | -0.010 |
| Fractures; n (%) | 44 (1.8%) | 52 (2.1%) | -0.0217 | 67 (1.4%) | 67 (1.4%) | 0.0000 | 111 (1.5%) | 119 (1.6%) | -0.008 |
| Falls v2; n (%) | 29 (1.2%) | 32 (1.3%) | -0.0090 | 28 (0.6%) | 26 (0.5%) | 0.0135 | 057 (0.8%) | 058 (0.8%) | 0.000 |
| Osteoporosis; n (%) | 63 (2.5%) | 56 (2.2%) | 0.0198 | 49 (1.0%) | 40 (0.8%) | 0.0212 | 112 (1.5%) | 096 (1.3%) | 0.017 |
| Depression; n (%) | 259 (10.4%) | 241 (9.6%) | 0.0267 | 320 (6.7%) | 321 (6.7%) | 0.0000 | 579 (7.9%) | 562 (7.7%) | 0.007 |
| Anxiety; n (%) | 323 (12.9%) | 318 (12.7%) | 0.0060 | 386 (8.0%) | 391 (8.1%) | -0.0037 | 709 (9.7%) | 709 (9.7%) | 0.000 |
| Sleep Disorder; n (%) | 153 (6.1%) | 148 (5.9%) | 0.0084 | 335 (7.0%) | 333 (6.9%) | 0.0039 | 488 (6.7%) | 481 (6.6%) | 0.004 |
| Dementia; n (%) | 34 (1.4%) | 25 (1.0%) | 0.0367 | 20 (0.4%) | 24 (0.5%) | -0.0149 | 054 (0.7%) | 049 (0.7%) | 0.000 |
| Delirium; n (%) | 19 (0.8%) | 19 (0.8%) | 0.0000 | 19 (0.4%) | 19 (0.4%) | 0.0000 | 038 (0.5%) | 038 (0.5%) | 0.000 |
| Psychosis; n (%) | 11 (0.4%) | 13 (0.5%) | -0.0149 | 17 (0.4%) | 13 (0.3%) | 0.0169 | 028 (0.4%) | 026 (0.4%) | 0.000 |
| Use of medications | | ì | | | | | | | |
| Use of ACE inhibitors; n (%) | 1,332 (53.3%) | 1,316 (52.7%) | 0.0120 | 2,689 (56.0%) | 2,716 (56.6%) | -0.0121 | 4,021 (55.1%) | 4,032 (55.2%) | -0.002 |
| Use of ARBs; n (%) | 486 (19.5%) | 498 (19.9%) | -0.0101 | 879 (18.3%) | 855 (17.8%) | 0.0130 | 1,365 (18.7%) | 1,353 (18.5%) | 0.005 |
| Use of Loop Diuretics - United; n (%) | 193 (7.7%) | 190 (7.6%) | 0.0038 | 254 (5.3%) | 286 (6.0%) | -0.0303 | 447 (6.1%) | 476 (6.5%) | -0.016 |
| Use of other diuretics- United; n (%) | 98 (3.9%) | 103 (4.1%) | -0.0102 | 188 (3.9%) | 207 (4.3%) | -0.0202 | 286 (3.9%) | 310 (4.2%) | -0.015 |
| Use of nitrates-United; n (%) | 1,089 (43.6%) | 1,086 (43.5%) | 0.0020 | 2,102 (43.8%) | 2,128 (44.3%) | -0.0101 | 3,191 (43.7%) | 3,214 (44.0%) | -0.006 |
| Use of other hypertension drugs; n (%) | 93 (3.7%) | 94 (3.8%) | -0.0053 | 150 (3.1%) | 163 (3.4%) | -0.0169 | 243 (3.3%) | 257 (3.5%) | -0.011 |
| Use of digoxin- United; n (%) | 21 (0.8%) | 20 (0.8%) | 0.0000 | 18 (0.4%) | 21 (0.4%) | 0.0000 | 039 (0.5%) | 041 (0.6%) | -0.014 |
| Use of Anti-arrhythmics; n (%) | 40 (1.6%) | 42 (1.7%) | -0.0079 | 73 (1.5%) | 74 (1.5%) | 0.0000 | 113 (1.5%) | 116 (1.6%) | -0.008 |
| Use of COPD/asthma meds- United; n (%) | 336 (13.5%) | 315 (12.6%) | 0.0267 | 529 (11.0%) | 526 (11.0%) | 0.0000 | 865 (11.8%) | 841 (11.5%) | 0.009 |
| Use of statins; n (%) | 2,267 (90.8%) | 2,280 (91.3%) | -0.0175 | 4,415 (91.9%) | 4,394 (91.5%) | 0.0145 | 6,682 (91.5%) | 6,674 (91.4%) | 0.004 |
| Use of other lipid-lowering drugs; n (%) | 179 (7.2%) | 189 (7.6%) | -0.0153 | 387 (8.1%) | 408 (8.5%) | -0.0145 | 566 (7.8%) | 597 (8.2%) | -0.015 |
| Use of antiplatelet agents; n (%) | 197 (7.9%) | 217 (8.7%) | -0.0290 | 322 (6.7%) | 359 (7.5%) | -0.0312 | 519 (7.1%) | 576 (7.9%) | -0.030 |
| Use of oral anticoagulants (Dabigatran, Rivaroxaban, Api | xa 56 (2.2%) | 58 (2.3%) | -0.0067 | 106 (2.2%) | 113 (2.4%) | -0.0133 | 162 (2.2%) | 171 (2.3%) | -0.007 |
| Use of heparin and other low-molecular weight heparins | ; ( 6 (0.2%) | 8 (0.3%) | -0.0200 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 006 (0.1%) | 008 (0.1%) | 0.000 |
| Use of NSAIDs; n (%) | 315 (12.6%) | 339 (13.6%) | -0.0296 | 700 (14.6%) | 702 (14.6%) | 0.0000 | 1,015 (13.9%) | 1,041 (14.3%) | -0.011 |
| Use of oral corticosteroids; n (%) | 386 (15.5%) | 372 (14.9%) | 0.0167 | 660 (13.7%) | 671 (14.0%) | -0.0087 | 1,046 (14.3%) | 1,043 (14.3%) | 0.000 |
| Use of bisphosphonate (United); n (%) | 25 (1.0%) | 22 (0.9%) | 0.0103 | 20 (0.4%) | 16 (0.3%) | 0.0169 | 045 (0.6%) | 038 (0.5%) | 0.014 |
| Use of opioids- United; n (%) | 540 (21.6%) | 533 (21.3%) | 0.0073 | 998 (20.8%) | 989 (20.6%) | 0.0049 | 1,538 (21.1%) | 1,522 (20.8%) | 0.007 |
| Use of antidepressants; n (%) | 421 (16.9%) | 409 (16.4%) | 0.0134 | 746 (15.5%) | 735 (15.3%) | 0.0055 | 1,167 (16.0%) | 1,144 (15.7%) | 0.008 |
| Use of antipsychotics; n (%) | 22 (0.9%) | 27 (1.1%) | -0.0201 | 36 (0.7%) | 45 (0.9%) | -0.0225 | 058 (0.8%) | 072 (1.0%) | -0.021 |
| Use of anticonvulsants; n (%) | 198 (7.9%) | 199 (8.0%) | -0.0037 | 286 (6.0%) | 296 (6.2%) | -0.0084 | 484 (6.6%) | 495 (6.8%) | -0.008 |
| Use of Benzos- United; n (%) | 249 (10.0%) | 247 (9.9%) | 0.0033 | 457 (9.5%) | 466 (9.7%) | -0.0068 | 706 (9.7%) | 713 (9.8%) | -0.003 |
| Use of anxiolytics/hypnotics- United; n (%) | 128 (5.1%) | 123 (4.9%) | 0.0092 | 242 (5.0%) | 240 (5.0%) | 0.0000 | 370 (5.1%) | 363 (5.0%) | 0.005 |
| Use of dementia meds- United; n (%) | 15 (0.6%) | 13 (0.5%) | 0.0135 | 5 (0.1%) | 7 (0.1%) | 0.0000 | 020 (0.3%) | 020 (0.3%) | 0.000 |
| Use of antiparkinsonian meds- United; n (%) | 27 (1.1%) | 31 (1.2%) | -0.0094 | 46 (1.0%) | 38 (0.8%) | 0.0212 | 073 (1.0%) | 069 (0.9%) | 0.010 |

| Use of glucose test strips; n (%) | 29 (1.2%) | 31 (1.2%) | 0.0000 | 58 (1.2%) | 60 (1.2%) | 0.0000 | 087 (1.2%) | 091 (1.2%) | 0.000 |
|---|---|---|---|---|---|---|---|---|---|
| Use of thiazide- United; n (%) | 192 (7.7%) | 188 (7.5%) | 0.0000 | 329 (6.9%) | 317 (6.6%) | 0.0120 | 521 (7.1%) | 505 (6.9%) | 0.008 |
| . , , | 2,164 (86.6%) | | 0.0073 | 4,241 (88.3%) | 4,252 (88.5%) | -0.0062 | 6,405 (87.7%) | 6,412 (87.8%) | -0.003 |
| Use of beta blockers; n (%) | <u> </u> | 2,160 (86.5%)<br>460 (18.4%) | 0.0029 | 780 (16.2%) | <u> </u> | -0.0082 | 1,242 (17.0%) | 1,263 (17.3%) | -0.003 |
| Use of calcium channel blockers; n (%) | 462 (18.5%) | <u> </u> | -0.0020 | <u> </u> | 803 (16.7%) | 0.0081 | 1,110 (15.2%) | 1,102 (15.1%) | 0.003 |
| Use of aspirin; n (%) | 312 (12.5%) | 320 (12.8%) | -0.0090 | 798 (16.6%) | 782 (16.3%) | 0.0081 | 1,894 (25.9%) | 1,890 (25.9%) | 0.000 |
| Use of Low Intensity Statins; n (%) | 626 (25.1%) | 633 (25.3%) | | 1,268 (26.4%) | 1,257 (26.2%) | | 5,571 (76.3%) | | 0.000 |
| Use of High Intensity Statins; n (%) | 1,910 (76.5%) | 1,892 (75.7%) | 0.0188 | 3,661 (76.2%) | 3,566 (74.3%) | 0.0440 | | 5,458 (74.8%) | -0.010 |
| Use of Sympatomimetic agents; n (%) | 27 (1.1%) | 31 (1.2%) | -0.0094 | 46 (1.0%) | 49 (1.0%) | 0.0000 | 073 (1.0%) | 080 (1.1%) | |
| Use of CNS stimulants; n (%) | 5 (0.2%) | 6 (0.2%) | 0.0000 | 27 (0.6%) | 27 (0.6%) | 0.0000 | 032 (0.4%) | 033 (0.5%) | -0.015 |
| All antidiabetic medications except Insulin; n (%) | 560 (22.4%) | 587 (23.5%) | -0.0262 | 1,099 (22.9%) | 1,109 (23.1%) | -0.0048 | 1,659 (22.7%) | 1,696 (23.2%) | -0.012 |
| DM Medications - Insulin Copy; n (%) | 217 (8.7%) | 219 (8.8%) | -0.0035 | 444 (9.2%) | 454 (9.5%) | -0.0103 | 661 (9.1%) | 673 (9.2%) | -0.003 |
| Use of estrogens, progestins, androgens; n (%) | 87 (3.5%) | 93 (3.7%) | -0.0107 | 210 (4.4%) | 216 (4.5%) | -0.0048 | 297 (4.1%) | 309 (4.2%) | -0.005 |
| Use of Angiogenesis inhibitors; n (%) | 1 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 001 (0.0%) | 000 (0.0%) | #DIV/0! |
| Use of Oral Immunosuppressants; n (%) | 3 (0.1%) | 3 (0.1%) | 0.0000 | 10 (0.2%) | 9 (0.2%) | 0.0000 | 013 (0.2%) | 012 (0.2%) | 0.000 |
| Use of fondaparinux or Bivalirudin; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 1 (0.0%) | #DIV/0! | 000 (0.0%) | 001 (0.0%) | #DIV/0! |
| Use of other direct thrombin inhibitors (lepirudin, desirud | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| Use of CYP inhibitors; n (%) | 406 (16.3%) | 407 (16.3%) | 0.0000 | 723 (15.1%) | 743 (15.5%) | -0.0111 | 1,129 (15.5%) | 1,150 (15.8%) | -0.008 |
| Use of CYP inducers; n (%) | 6 (0.2%) | 8 (0.3%) | -0.0200 | 19 (0.4%) | 16 (0.3%) | 0.0169 | 025 (0.3%) | 024 (0.3%) | 0.000 |
| Burden of disease/Healthcare utilization | | | | | | | | | |
| Combined comorbidity score, 180 days Copy | | | | | | | | | |
| mean (sd) | 1.19 (1.81) | 1.21 (1.83) | -0.0110 | 0.60 (1.47) | 0.61 (1.47) | -0.0068 | 0.80 (1.59) | 0.82 (1.60) | -0.013 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.0000 | 0.00 [-1.00, 1.00] | 0.00 [-1.00, 1.00] | 0.0000 | 0.34 (1.59) | 0.34 (1.60) | 0.000 |
| Frailty Score (mean): Empirical Version 365 days, v2 | | | | | | | | | |
| mean (sd) | 0.18 (0.04) | 0.18 (0.04) | 0.0000 | 0.17 (0.03) | 0.17 (0.03) | 0.0000 | 0.17 (0.03) | 0.17 (0.03) | 0.000 |
| median [IQR] | 0.17 [0.15, 0.20] | 0.17 [0.15, 0.20] | 0.0000 | 0.16 [0.14, 0.18] | 0.16 [0.15, 0.18] | 0.0000 | 0.16 (0.03) | 0.16 (0.03) | 0.000 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd digit level | | | | | | | | | |
| mean (sd) | 8.40 (8.59) | 8.76 (8.97) | -0.0410 | 6.01 (7.71) | 6.05 (7.67) | -0.0052 | 6.83 (8.02) | 6.98 (8.14) | -0.019 |
| median [IQR] | 7.00 [0.00, 14.00] | 8.00 [0.00, 14.00] | -0.1139 | 0.00 [0.00, 12.00] | 0.00 [0.00, 12.00] | 0.0000 | 2.40 (8.02) | 2.74 (8.14) | -0.042 |
| HAS-BLED Score (ICD-9 and ICD-10), 180 days | | | | | | | | | |
| mean (sd) | 3.43 (0.57) | 3.43 (0.58) | 0.0000 | 3.16 (0.46) | 3.15 (0.45) | 0.0220 | 3.25 (0.50) | 3.25 (0.50) | 0.000 |
| median [IQR] | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.0000 | 3.00 [3.00, 3.00] | 3.00 [3.00, 3.00] | 0.0000 | 3.00 (0.50) | 3.00 (0.50) | 0.000 |
| number of different/distinct medication prescriptions | | | | | | | | | |
| mean (sd) | 8.75 (4.38) | 8.77 (4.50) | -0.0045 | 8.58 (4.15) | 8.63 (4.23) | -0.0119 | 8.64 (4.23) | 8.68 (4.32) | -0.009 |
| median [IQR] | 8.00 [6.00, 11.00] | 8.00 [5.00, 11.00] | 0.0000 | 8.00 [6.00, 11.00] | 8.00 [6.00, 11.00] | 0.0000 | 8.00 (4.23) | 8.00 (4.32) | 0.000 |
| Any hospitalization within prior 30 days; n (%) | 2,498 (100.0%) | 2,498 (100.0%) | #DIV/0! | 4,802 (100.0%) | 4,802 (100.0%) | #DIV/0! | 7,300 (100.0%) | 7,300 (100.0%) | #DIV/0! |
| Number of Hospitalizations | | | | | | | | | |
| mean (sd) | 1.08 (0.30) | 1.08 (0.32) | 0.0000 | 1.06 (0.28) | 1.06 (0.26) | 0.0000 | 1.07 (0.29) | 1.07 (0.28) | 0.000 |
| median [IQR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.0000 | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.0000 | 1.00 (0.29) | 1.00 (0.28) | 0.000 |
| Number of hospital days | | | | | | | | | |
| mean (sd) | 3.61 (1.95) | 3.60 (2.15) | 0.0049 | 3.48 (2.00) | 3.50 (1.64) | -0.0109 | 3.52 (1.98) | 3.53 (1.83) | -0.005 |
| median [IQR] | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.0000 | 3.00 [3.00, 4.00] | 3.00 [3.00, 4.00] | 0.0000 | 3.00 (1.98) | 3.00 (1.83) | 0.000 |
| Number of Emergency Department (ED) visits v3 | | | | | | | | | |
| mean (sd) | 1.09 (1.26) | 1.10 (1.37) | -0.0076 | 3.59 (5.64) | 3.62 (6.71) | -0.0048 | 2.73 (4.63) | 2.76 (5.50) | -0.006 |
| median [IQR] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.0000 | 2.00 [0.00, 4.00] | 2.00 [0.00, 4.00] | 0.0000 | 1.66 (4.63) | 1.66 (5.50) | 0.000 |
| Number of Office visits | | | | | | | | | |
| mean (sd) | 2.98 (3.14) | 3.03 (3.30) | -0.0155 | 2.69 (2.85) | 2.70 (2.91) | -0.0035 | 2.79 (2.95) | 2.81 (3.05) | -0.007 |
| median [IQR] | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 0.0000 | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 0.0000 | 2.00 (2.95) | 2.00 (3.05) | 0.000 |
| Number of internal medicine/family medicine visits | | | | | | | | | |
| mean (sd) | 6.26 (8.89) | 6.47 (10.55) | -0.0215 | 3.83 (5.90) | 3.86 (6.58) | -0.0048 | 4.66 (7.07) | 4.75 (8.16) | -0.012 |
| median [IQR] | 3.00 [1.00, 8.00] | 3.00 [1.00, 8.00] | 0.0000 | 2.00 [0.00, 5.00] | 2.00 [0.00, 5.00] | 0.0000 | 2.34 (7.07) | 2.34 (8.16) | 0.000 |
| Number of Cardiologist visits | | | | | | | | | |

| mean (sd) | 8.18 (5.00) | 8.14 (5.05) | 0.0080 | 1.00 (2.09) | 1.02 (2.27) | -0.0092 | 3.46 (3.38) | 3.46 (3.48) | 0.000 |
|---|---|---|---|---|---|---|---|---|---|
| median [IQR] | 8.00 [5.00, 11.00] | 7.00 [5.00, 10.00] | 0.1990 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.0000 | 2.74 (3.38) | 2.40 (3.48) | 0.099 |
| Number electrocardiograms received v2 | | , , , , , , | | , , , , , , | | | , , | , , | |
| mean (sd) | 3.33 (2.45) | 3.33 (2.62) | 0.0000 | 0.97 (1.32) | 0.97 (1.36) | 0.0000 | 1.78 (1.79) | 1.78 (1.89) | 0.000 |
| median [IQR] | 3.00 [2.00, 4.00] | 3.00 [2.00, 5.00] | 0.0000 | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.0000 | 1.68 (1.79) | 1.68 (1.89) | 0.000 |
| Number of BNP tests | | | | | | | ` ' | , , | |
| mean (sd) | 0.11 (0.37) | 0.10 (0.40) | 0.0260 | 0.12 (0.37) | 0.12 (0.38) | 0.0000 | 0.12 (0.37) | 0.11 (0.39) | 0.026 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.37) | 0.00 (0.39) | 0.000 |
| Number of Cardiac biomarkers tests (tropnin, CK-MBs, My | | [0.00, 0.00] | | [,] | [,] | | ( , | | |
| mean (sd) | 0.68 (1.63) | 0.73 (1.73) | -0.0297 | 0.72 (1.67) | 0.73 (1.60) | -0.0061 | 0.71 (1.66) | 0.73 (1.65) | -0.012 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.00 (1.66) | 0.00 (1.65) | 0.000 |
| Number of Ambulatory Blood pressure monitoring tests | 0.00 [0.00) | 0.00 [0.00) 2.00] | | 0.00 [0.00) 2.00] | 0.00 [0.00, 2.00] | | , | | |
| mean (sd) | 0.00 (0.03) | 0.00 (0.02) | 0.0000 | 0.00 (0.04) | 0.00 (0.03) | 0.0000 | 0.00 (0.04) | 0.00 (0.03) | 0.000 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.04) | 0.00 (0.03) | 0.000 |
| N of days on antihypertensive medications during baseline | | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.0.1) | 0.00 (0.00) | 0.000 |
| mean (sd) | 75.35 (78.69) | 75.92 (78.36) | -0.0073 | 71.06 (77.53) | 71.15 (77.62) | -0.0012 | 72.53 (77.93) | 72.78 (77.87) | -0.003 |
| median [IQR] | | 35.00 [1.00, 168.00] | -0.0509 | | 12.00 [1.00, 164.00] | 0.0258 | 19.82 (77.93) | 19.87 (77.87) | -0.001 |
| N of days in database anytime prior | 52.55 [1.55, 105.00] | 55.00 [1.00, 100.00] | 0.0303 | [1.00, 100.00] | 00 [1.00, 104.00] | 0.0250 | 25.52 (77.55) | 25.0. (11.01) | 0.001 |
| mean (sd) | 1,658.31 (1,306.21) | 1,660.85 (1,331.74) | -0.0019 | 1,989.48 (1,379.50) | 1 998 92 (1 372 00) | -0.0069 | 1876.16 (1354.87) | 1883.24 (1358.36) | -0.005 |
| median [IQR] | | 41,227.50 [593.75, 2,4 | 0.0140 | | 1,693.00 [824.75, 3,0 | -0.0076 | 1533.13 (1354.87) | 1533.71 (1358.36) | 0.000 |
| Mean Copay for per prescription cost (charges in U.S. \$) (3 | | 1,227.30 [333.73, 2,4 | 0.01.0 | 1,002.30 [000.00, 3,0 | 1,055.00 [024.75, 5,0 | 0.0070 | 1555115 (155 1167) | 1555171 (1555150) | 0.000 |
| mean (sd) | 23.00 (28.64) | 23.95 (28.18) | -0.0334 | 16.82 (22.87) | 16.49 (20.73) | 0.0151 | 18.93 (24.99) | 19.04 (23.55) | -0.005 |
| median [IQR] | 14.98 [6.00, 29.47] | 15.31 [6.44, 30.82] | -0.0116 | 10.69 [2.63, 22.50] | 10.42 [2.98, 22.00] | 0.0131 | 12.16 (24.99) | 12.09 (23.55) | 0.003 |
| | 351 (14.1%) | 361 (14.5%) | -0.0114 | 739 (15.4%) | 743 (15.5%) | -0.0028 | 1,090 (14.9%) | 1,104 (15.1%) | -0.006 |
| Missing; n (%) Duration of index hospitalization (i.e. anchor hospitalization | <del></del> | 301 (14.3%) | -0.0114 | 739 (13.4%) | 743 (15.5%) | -0.0028 | 1,090 (14.970) | 1,104 (13.170) | -0.000 |
| mean (sd) | 1.00 (0.00) | 1.00 (0.00) | #DIV/0! | 1.00 (0.00) | 1.00 (0.00) | #DIV/0! | 1.00 (0.00) | 1.00 (0.00) | #DIV/0! |
| | 1.00 (0.00) | 1.00 (0.00) | #DIV/0! | 1.00 (0.00) | 1.00 (0.00) | #DIV/0! | 1.00 (0.00) | 1.00 (0.00) | #DIV/0! |
| median [IQR] N of Generic name drugs | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | #DIV/U: | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | #DIV/U: | 1.00 (0.00) | 1.00 (0.00) | #DIV/0: |
| mean (sd) | 12.43 (11.07) | 12.50 (11.04) | -0.0063 | 10.82 (9.17) | 10.89 (9.29) | -0.0076 | 11.37 (9.86) | 11.44 (9.92) | -0.007 |
| | | | 0.0000 | 8.00 [4.00, 14.00] | | 0.0000 | 8.34 (9.86) | 8.34 (9.92) | 0.000 |
| median [IQR] N of Brand name drugs | 9.00 [5.00, 16.00] | 9.00 [5.00, 16.00] | 0.0000 | 8.00 [4.00, 14.00] | 8.00 [4.00, 14.00] | 0.0000 | 8.54 (3.80) | 8.54 (3.32) | 0.000 |
| | 3.15 (3.47) | 3.17 (4.09) | -0.0053 | 3.53 (3.65) | 3.59 (3.74) | -0.0162 | 3.40 (3.59) | 3.45 (3.86) | -0.013 |
| mean (sd)<br>median [IQR] | | 2.00 [1.00, 4.00] | 0.0000 | 2.00 [1.00, 4.00] | | 0.0000 | 2.00 (3.59) | 2.00 (3.86) | 0.000 |
| | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 0.0000 | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 0.0000 | 2.00 (3.39) | 2.00 (3.80) | 0.000 |
| Number of D-dimer tests | 0.00 (0.30) | 0.00 (0.30) | 0.0000 | 0.07 (0.30) | 0.07 (0.28) | 0.0000 | 0.07 (0.29) | 0.07 (0.27) | 0.000 |
| mean (sd) | 0.06 (0.26)<br>0.00 [0.00, 0.00] | 0.06 (0.26)<br>0.00 [0.00, 0.00] | 0.0000 | 0.07 (0.30)<br>0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.29) | 0.00 (0.27) | 0.000 |
| median [IQR] Numbe of CRP, high-sensitivity CRP tests | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.29) | 0.00 (0.27) | 0.000 |
| mean (sd) | 0.05 (0.27) | 0.04 (0.24) | 0.0391 | 0.04 (0.25) | 0.04 (0.24) | 0.0000 | 0.04 (0.26) | 0.04 (0.24) | 0.000 |
| | | | 0.0000 | 0.04 (0.23) | | 0.0000 | 0.00 (0.26) | 0.00 (0.24) | 0.000 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (0.20) | 0.00 (0.24) | 0.000 |
| Number of PT or aPTTt tests | 0.27 (1.05) | 0.27 (1.00) | 0.0000 | 0.20 (0.08) | 0.40 (1.03) | -0.0100 | 0.38 (1.00) | 0.39 (1.01) | -0.010 |
| mean (sd) | 0.37 (1.05) | 0.37 (1.00) | | 0.39 (0.98) | 0.40 (1.02) | | ` ' | 0.00 (1.01) | |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (1.00) | 0.00 (1.01) | 0.000 |
| Number of Bleeding time tests | 0.00 (0.00) | 0.00 (0.00) | #DIV/OI | 0.00 (0.00) | 0.00 (0.00) | #DIV/01 | 0.00 (0.00) | 0.00 (0.00) | #DIV/0! |
| mean (sd) | (00.0) (00.0) | 0.00 (0.00) | #DIV/0! | (00.0) (00.0) | (00.0) (00.0) | #DIV/0! | 0.00 (0.00) | 0.00 (0.00) | |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | #DIV/0! | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | #DIV/0! | | | #DIV/0! |
| Occurrence of creatinine tests ordered (for PS); n (%) | 68 (2.7%) | 68 (2.7%) | 0.0000 | 119 (2.5%) | 130 (2.7%) | -0.0126 | 187 (2.6%) | 198 (2.7%) | -0.006 |
| Cardiovascular stress test; n (%) | 8 (0.3%) | 5 (0.2%) | 0.0200 | 10 (0.2%) | 10 (0.2%) | 0.0000 | 018 (0.2%) | 015 (0.2%) | 0.000 |
| Echocardiogram; n (%) | 1,774 (71.0%) | 1,764 (70.6%) | 0.0088 | 3,228 (67.2%) | 3,232 (67.3%) | -0.0021 | 5,002 (68.5%) | 4,996 (68.4%) | 0.002 |
| Colonoscopy; n (%) | 79 (3.2%) | 84 (3.4%) | -0.0112 | 178 (3.7%) | 177 (3.7%) | 0.0000 | 257 (3.5%) | 261 (3.6%) | -0.005 |
| Fecal occult blood (FOB) test; n (%) | 67 (2.7%) | 69 (2.8%) | -0.0061 | 114 (2.4%) | 116 (2.4%) | 0.0000 | 181 (2.5%) | 185 (2.5%) | 0.000 |
| Flu vaccine; n (%) | 348 (13.9%) | 337 (13.5%) | 0.0116 | 412 (8.6%) | 404 (8.4%) | 0.0072 | 760 (10.4%) | 741 (10.2%) | 0.007 |

| Mammogram; n (%) | 116 (4.6%) | 120 (4.8%) | -0.0095 | 156 (3.2%) | 168 (3.5%) | -0.0167 | 272 (3.7%) | 288 (3.9%) | -0.010 |
|---|---|---|---|---|---|---|---|---|---|
| Pap smear; n (%) | 49 (2.0%) | 49 (2.0%) | 0.0000 | 100 (2.1%) | 96 (2.0%) | 0.0071 | 149 (2.0%) | 145 (2.0%) | 0.000 |
| Pneumonia vaccine; n (%) | 377 (15.1%) | 400 (16.0%) | -0.0248 | 343 (7.1%) | 331 (6.9%) | 0.0078 | 720 (9.9%) | 731 (10.0%) | -0.003 |
| PSA test or Prostate exam for DRE; n (%) | 380 (15.2%) | 385 (15.4%) | -0.0056 | 621 (12.9%) | 632 (13.2%) | -0.0089 | 1,001 (13.7%) | 1,017 (13.9%) | -0.006 |
| Bone mineral density; n (%) | 39 (1.6%) | 41 (1.6%) | 0.0000 | 34 (0.7%) | 32 (0.7%) | 0.0000 | 073 (1.0%) | 073 (1.0%) | 0.000 |
| Drug eluting stent; n (%) | 826 (33.1%) | 800 (32.0%) | 0.0235 | 1,804 (37.6%) | 1,804 (37.6%) | 0.0000 | 2,630 (36.0%) | 2,604 (35.7%) | 0.006 |
| Bare metal stent; n (%) | 2,143 (85.8%) | 2,146 (85.9%) | -0.0029 | 3,978 (82.8%) | 3,958 (82.4%) | 0.0106 | 6,121 (83.8%) | 6,104 (83.6%) | 0.005 |